CLINICAL TRIAL: NCT01774786
Title: A Double-Blind, Placebo-Controlled, Randomized, Multicenter Phase III Study Evaluating the Efficacy and Safety of Pertuzumab in Combination With Trastuzumab and Chemotherapy in Patients With HER2-Positive Metastatic Gastroesophageal Junction and Gastric Cancer
Brief Title: A Study of Pertuzumab in Combination With Trastuzumab and Chemotherapy in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Gastroesophageal Junction or Gastric Cancer
Acronym: JACOB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO25114; 2012-003554-83 (EudraCT Number)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Capecitabine; Cisplatin; pertuzumab; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pertuzumab + Trastuzumab + Chemotherapy (Experimental): Participants will receive pertuzumab in combination with trastuzumab and chemotherapy (cisplatin and fluoropyrimidine [capecitabine or 5-fluorouracil]) for the first 6 treatment cycles (cycle length = 21 days). Thereafter, participants will continue to receive pertuzumab and trastuzumab until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Interventions: Drug: 5-Fluorouracil; Drug: Capecitabine; Drug: Cisplatin; Drug: Pertuzumab; Drug: Trastuzumab
- Placebo + Trastuzumab + Chemotherapy (Placebo Comparator): Participants will receive placebo in combination with trastuzumab and chemotherapy (cisplatin and fluoropyrimidine [capecitabine or 5-fluorouracil]) for the first 6 treatment cycles (cycle length = 21 days). Thereafter, participants will continue to receive placebo and trastuzumab until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Interventions: Drug: 5-Fluorouracil; Drug: Capecitabine; Drug: Cisplatin; Drug: Placebo; Drug: Trastuzumab

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive 5-fluorouracil 800 milligrams per meter square (mg/m^2)/24 hour IV infusion for 120 hours (Days 1-5) q3w for 6 cycles.
Drug: Capecitabine — Participants will receive capecitabine 1000 mg/m^2 orally twice daily, evening of Day 1 to morning of Day 15 (28 doses) q3w for 6 cycles.
  Other Names: Xeloda
Drug: Cisplatin — Participants will receive cisplatin 80 mg/m^2 IV q3w for 6 cycles.
Drug: Pertuzumab — Participants will receive pertuzumab 840 mg IV q3w until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Other Names: Perjeta; RO4368451
  Arms: Pertuzumab + Trastuzumab + Chemotherapy
Drug: Placebo — Participants will receive placebo (matched to pertuzumab) IV q3w until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Arms: Placebo + Trastuzumab + Chemotherapy
Drug: Trastuzumab — Participants will receive 8 mg/kg IV initial dose on Day 1, followed by 6 mg/kg IV q3w until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Other Names: Herceptin; RO0452317

SUMMARY:
This double-blind, placebo-controlled, randomized, multicenter, international, parallel arm study will evaluate the efficacy and safety of pertuzumab in combination with trastuzumab, fluoropyrimidine and cisplatin as first-line treatment in participants with HER2-positive metastatic gastroesophageal junction (GEJ) or gastric cancer (GC). Participants will be randomized to receive pertuzumab 840 milligrams (mg) or placebo intravenously every 3 weeks (q3w) in combination with trastuzumab (initial dose of 8 milligrams per kilogram [mg/kg] intravenously [IV] followed by 6 mg/kg IV q3w) and cisplatin and fluoropyrimidine (capecitabine or 5-fluorouracil) for the first 6 treatment cycles. Participants will continue to receive pertuzumab or placebo and trastuzumab until disease progression occurrence of unacceptable toxicity or withdrawal from the study for another reason.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the stomach or GEJ
* Measurable or evaluable non-measurable disease as assessed by the investigator according to RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy greater than equal to (>/=) 3 months

Exclusion Criteria:

* Previous cytotoxic chemotherapy for advanced (metastatic) disease
* Evidence of disease progression documented within 6 months after completion of prior neoadjuvant or adjuvant cytotoxic chemotherapy, or both, or radiotherapy for GEJ adenocarcinoma
* Previous treatment with any HER2-directed therapy, at any time, for any duration
* Previous exposure to any investigational treatment within 30 days before the first dose of study treatment
* Radiotherapy within 30 days before the first dose of study treatment (within 2 weeks if given as palliation to bone metastases, if recovered from all toxicities)
* History or evidence of brain metastases
* Clinically significant active gastrointestinal (GI) bleeding (Grade >/=2 according to National Cancer Institute [NIC]-Common Terminology Criteria for Adverse Events Version 4.0 [CTCAEv.4.0])
* Residual toxicity resulting from previous therapy (for example, hematologic, cardiovascular, or neurologic toxicity that is Grade >/=2). Alopecia is permitted
* Other malignancy (in addition to gastric cancer [GC]) within 5 years before enrollment, except for carcinoma in situ of the cervix or squamous or basal cell carcinoma of the skin that has been previously treated with curative intent
* Inadequate hematologic, renal or liver function
* Pregnant or lactating women
* History of congestive heart failure of any New York Heart Association (NYHA) criteria
* Angina pectoris requiring treatment
* Myocardial infarction within the past 6 months before the first dose of study drug
* Clinically significant valvular heart disease or uncontrollable high-risk cardiac arrhythmia
* History or evidence of poorly controlled hypertension
* Baseline left ventricular ejection fraction (LVEF) value less than (<) 55 percent (%)
* Any significant uncontrolled intercurrent systemic illness
* Positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (172):
- United States (10):
  - Florida Cancer Specialists - SCRI; Pharmacy, Fort Myers, Florida
  - University Of Chicago Medical Center; Section Of Hematology/Oncology, Chicago, Illinois
  - Indiana University Health; Goshen Center for Cancer Care, Goshen, Indiana
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Queens Medical Associates, Fresh Meadows, New York
  - Weill Medical College of Cornell University; Division of Hematology & Medical Oncology, New York, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Medical University of South Carolina; Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology PLLC - Nashville (20th Ave), Nashville, Tennessee
- Australia (4):
  - Royal Brisbane Womens Hosp; Division of Oncology, Herston, Queensland
  - Monash Medical Centre; Oncology, Clayton, Victoria
  - Austin Health; Cancer Clinical Trial Centre, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital; Medical Oncology, Perth, Western Australia
- Austria (2):
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Krankenhaus St. Vinzenz Der Barmherzigen Schwestern Zams; Abt. Für Innere Medizin, Zams
- Cliniques Universitaires St-Luc, Brussels, Belgium
- Brazil (8):
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Clinica de Oncologia Medica, São Paulo, São Paulo
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP*X, São Paulo, São Paulo
- Bulgaria (3):
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - MHAT Serdika, Sofia
  - SHATOD Dr. Marko Antonov Markov-Varna, EOOD; Department of Medicinall Onchotherapy and Palliative, Varna
- Canada (7):
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Toronto East General Hospital; Haematology/Oncology, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Mount Sinai Hospital; Oncology, Toronto, Ontario
  - McGill University; Glen Site; Oncology, Montreal, Quebec
- China (22):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Changzhou First People's Hospital, Changzhou
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - Fuzhou General Hospital, PLA Nanjing Military Area Command, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - The 81st Hospital of P.L.A., Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - General Hospital of Shenyang Military Command of PLA, Shenyang
  - Hebei Medical University Fourth Hospital;(Tumor Hospital of Hebei Province), Shijiazhuang
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Croatia (2):
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Sisters of Mercy, Zagreb
- Hospital Oncologia; Oncology, San Salvador, El Salvador
- Finland (2):
  - Docrates Cance Center, Helsinki
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- Germany (11):
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - Kliniken Essen-Mitte, Evang. Huyssens-Stiftung, Klinik für Internistische Onkologie / Haematologie, Essen
  - Klinik Esslingen; Klinik für Allgemeine Innere Medizin, Onkologie/Haematologie, Esslingen am Neckar
  - Universitätsklinikum Hamburg-Eppendorf; Hubertus Wald Tumorzentrum, Hamburg
  - Universitaetsklinikum Leipzig, Universitaeres Krebszentrum Leipzig (UCCL), Leipzig
  - Klinikum Ludwigsburg; Studiensekretariat, Ludwigsburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz; II. Medizinische Klinik, Mainz
  - Universitätsklinikum Mannheim, Tagestherapiezentrum, Interdisziplinäres Tumorzentrum, Mannheim
  - Philipps-Universität Marburg; Klinik für Innere Med.; Schwerpunkt Hämatologie/Onkologie/Immunologie, Marburg
  - Universitätsklinikum Ulm; Zentrum für Innere Medizin Klinik für Innere Medizin I, Ulm
- Medical Solution; Hematology, Guatemala City, Guatemala
- Hungary (5):
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Onkologiai Klinika, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz;Sugarterapias Klinikai Onkologiai Intez, Miskolc
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Italy (12):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Seconda Universita' Degli Studi; Divsione Di Oncologia Medica, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - AUSL - IRCCS Santa Maria Nuova; U.O. Day Hospital di Oncologia, Reggio Emilia, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Ospedali Riuniti Di Ancona; Oncology, Ancona, The Marches
  - Azlenda Ospendaliero-Universitaria Pisana; C.O. Oncologia 2, Pisa, Tuscany
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
- Japan (15):
  - Aichi Cancer Center Hospital; Clinical Oncology, Aichi
  - Nagoya university Hospital; Gastroenterological Surgery 2, Aichi
  - National Cancer Center Hospital East; Gastroenterology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Gastroenterology, Ehime
  - Kyushu University Hospital; Surgery and Science, Fukuoka
  - Gifu University Hospital; Digestive Surgery, Gifu
  - Hiroshima City Hiroshima Citizens Hospital; Surgery, Hiroshima
  - Kobe city Medical center General Hospital; Medical Oncology, Hyōgo
  - St.Marianna University School of Medicine hospital; Medical Oncology, Kanagawa
  - Kanagawa Cancer Center; Gastrointestinal Surgery, Kanagawa
  - Osaka International Cancer Institute;; Medical oncology and Gastrointestinal oncology, Osaka
  - Osaka General Medical Center; Gastroenterological Surgery, Osaka
  - Saitama Cancer Center; Gastroenterology, Saitama
  - National Cancer Center Hospital; Gastrointestinal Oncology, Tokyo
  - Toyama University Hospital;Gastroenterology and Hematology, Toyama
- Kazakh Scientific Research Institution Of Oncology and Radiology; Chemotherapy department, Almaty, Kazakhstan
- Malaysia (4):
  - Hospital Universiti Sains Malaysia [Neurology], Kubang Kerian, Kelantan
  - Hospital Wanita dan Kanak-Kanak Sabah, Sabah, Sabah
  - Hospital Kuala Lumpur; Jabatan Radioterapi dan Onkologi, Kuala Lumpur
  - University Malaya Medical Centre; Clinical Oncology Unit,, Kuala Lumpur
- Mexico (3):
  - Hospital Angeles Metropolitano; Room 220, Mexico City, Mexico CITY (federal District)
  - Inst. Nacional de Cancerologia; Investigacion Clinica, Mexico City
  - Oaxaca Site Management Organization, Oaxaca City
- Academisch Medisch Centrum Universiteit Amsterdam, Amsterdam, Netherlands
- North Macedonia (2):
  - Clinical Hospital; Oncology Department, Bitola
  - University Clinic for Radiotherapy and Oncology, Skopje
- Medical Research Centre, Panama City, Panama
- Peru (5):
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital Sabogal; Oncology, Callao
  - Hosp Nacion Edgardo Rebagliati; Oncologia Medica, Jesus Maria
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Clinica San Borja, Lima
- Poland (8):
  - Bialostockie Ctr Onkologii; Oddzial Chemioterapii Dziennej, Bialystok
  - Szpital Specjalistyczny Podkarpacki Ośrodek Onkologiczny, Brzozów
  - Centrum Onkologii;Im. Franciszka Lukaszczyka;Onkologii, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - SPZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarawskiego, Opole
  - NZOZ Centrum Medyczne HCP Sp. z o.o., Poznan
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie; Klinika Gastroenterologii Onkologicznej, Warsaw
- Romania (3):
  - Cardiomed Medical Center, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Euroclinic Center of Oncology SRL, Iași
- Russia (4):
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - Clinical Oncology Dispensary; Chemotherapy, Omsk
  - SBI for HPE "Ryazan State Medical University n.a. I.P. Pavlov" of MoH of RF, Ryazan
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
- South Korea (6):
  - Kyungpook National University Medical Center, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei Medical Center; Dept. of Medicine , Division of Hemato-Oncology, Seoul
  - Asan Medical Center; Medical Oncology, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (9):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
- Switzerland (2):
  - CHUV; Departement d'Oncologie, Lausanne
  - Luzerner Kantonsspital; Medizinische Onkologie, Lucerne
- Taiwan (5):
  - Taichung Veterans General Hospital; Dept of Surgery, Taichung
  - National Cheng Kung University Hospital; Oncology, Tainan
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- Thailand (5):
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Khonkaen Hospital, Khonkaen
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Turkey (Türkiye) (7):
  - Ankara Uni School of Medicine; Medical Oncology, Ankara
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - TC Necmettin Erbakan University Meram Medical Faculty Hospital, Konya
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya

REFERENCES:
- [Derived] Tabernero J, Hoff PM, Shen L, Ohtsu A, Shah MA, Siddiqui A, Heeson S, Kiermaier A, Macharia H, Restuccia E, Kang YK. Pertuzumab, trastuzumab, and chemotherapy in HER2-positive gastric/gastroesophageal junction cancer: end-of-study analysis of the JACOB phase III randomized clinical trial. Gastric Cancer. 2023 Jan;26(1):123-131. doi: 10.1007/s10120-022-01335-4. Epub 2022 Sep 6. PMID 36066725
- [Derived] Liu T, Qin Y, Li J, Xu R, Xu J, Yang S, Qin S, Bai Y, Wu C, Mao Y, Wu H, Ge Y, Shen L. Pertuzumab in combination with trastuzumab and chemotherapy for Chinese patients with HER2-positive metastatic gastric or gastroesophageal junction cancer: a subpopulation analysis of the JACOB trial. Cancer Commun (Lond). 2019 Jun 24;39(1):38. doi: 10.1186/s40880-019-0384-6. PMID 31234927
- [Derived] Kirschbrown WP, Wang B, Nijem I, Ohtsu A, Hoff PM, Shah MA, Shen L, Kang YK, Alsina M, Girish S, Garg A. Pharmacokinetic and exposure-response analysis of pertuzumab in patients with HER2-positive metastatic gastric or gastroesophageal junction cancer. Cancer Chemother Pharmacol. 2019 Sep;84(3):539-550. doi: 10.1007/s00280-019-03871-w. Epub 2019 Jun 10. PMID 31183514
- [Derived] Tabernero J, Hoff PM, Shen L, Ohtsu A, Shah MA, Cheng K, Song C, Wu H, Eng-Wong J, Kim K, Kang YK. Pertuzumab plus trastuzumab and chemotherapy for HER2-positive metastatic gastric or gastro-oesophageal junction cancer (JACOB): final analysis of a double-blind, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2018 Oct;19(10):1372-1384. doi: 10.1016/S1470-2045(18)30481-9. Epub 2018 Sep 11. PMID 30217672

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 780 participants were enrolled in the study.
Groups:
- Pertuzumab + Trastuzumab + Chemotherapy: Participants received pertuzumab in combination with trastuzumab and chemotherapy (cisplatin and fluoropyrimidine [capecitabine or 5-fluorouracil]) for the first 6 treatment cycles (cycle length = 21 days). Thereafter, participants continued to receive pertuzumab and trastuzumab until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
- Placebo + Trastuzumab + Chemotherapy: Participants received placebo in combination with trastuzumab and chemotherapy (cisplatin and fluoropyrimidine [capecitabine or 5-fluorouracil]) for the first 6 treatment cycles (cycle length = 21 days). Thereafter, participants continued to receive placebo and trastuzumab until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Started (Intent-to-Treat (ITT) population) | 388 | 392
Did Not Receive Any Study Treatment | 4 (2 patients found ineligible after enrollment and 2 patients died before treatment.) | 3 (All 3 patients found ineligible for the study after enrollment and before treatment.)
Received at Least One Dose of Pertuzumab (Pertuzumab Safety Population) | 384 | 1 (One participant randomized to placebo arm received 1 dose of pertuzumab by error.)
Received Placebo (No Pertuzumab) (Placebo Safety Population) | 0 | 388
Completed | 60 | 46
Not Completed | 328 | 346
Not completed — Death | 300 | 319
Not completed — Lost to Follow-up | 6 | 7
Not completed — Withdrawal by Subject | 18 | 14
Not completed — Physician Decision | 2 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Reason Not Specified | 2 | 5

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants regardless of whether treatment was actually received, with participants grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy | Total
Number analyzed (Participants) | 388 | 392 | 780
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.3) | 60.1 (10.7) | 60.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 69 | 163
  Male | 294 | 323 | 617
Geographic Region [Count of Participants; unit: Participants] — Participants were stratified at randomization according to geographic region, prior gastrectomy, and HER2 status.
  Participants
    Asia (excluding Japan) | 143 | 146 | 289
    Japan | 40 | 40 | 80
    North America/Western Europe/Australia | 133 | 133 | 266
    South America/Eastern Europe | 72 | 73 | 145
Prior Gastrectomy [Count of Participants; unit: Participants] — Participants were stratified at randomization according to geographic region, prior gastrectomy, and HER2 status.
  Participants
    Prior Gastrectomy | 105 | 102 | 207
    No Prior Gastrectomy | 283 | 290 | 573
Human Epidermal Growth Factor Receptor 2 (HER2) Status [Count of Participants; unit: Participants] — Participants were stratified at randomization according to geographic region, prior gastrectomy, and HER2 status. HER2 positivity of tumor specimens from each participant were determined by central laboratory testing. The IHC gives a score of 0 to 3+ that measures the amount of HER2 proteins on the surface of cells. A participant's cancer was considered HER2-positive with an IHC score of 2+ that was confirmed by ISH positivity or by an IHC score of 3+. IHC = immunohistochemistry; ISH = in-situ hybridization
  Participants
    IHC 2+/ISH+ | 129 | 130 | 259
    IHC 3+ | 259 | 262 | 521
Measurability of Disease, per RECIST v1.1 [Count of Participants; unit: Participants]
  Measurable Disease | 351 | 352 | 703
  Non-Measurable Evaluable Disease Only | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. For participants who were still alive on the date of clinical data cut-off for the OS analysis, the last date when the participant was known to be alive on, or prior to the clinical cut-off date, was used to determine the censoring date. Participants who did not have any post-baseline data (e.g., dosing records, imaging dates, visit dates) were censored at the date of randomization plus 1 day.
Time Frame: From Baseline until death from any cause (Median [full range] duration of follow-up in Pertuzumab vs. Placebo arms for Primary Analysis: 24.4 [0-42] months vs. 25.0 [0-41] months; Final Analysis: 46.1 [0-70] months vs. 44.4 [0-68] months)
Population: The intent-to-treat (ITT) population included all randomized participants, regardless of whether study medication was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 388 | 392
Months
  Primary Analysis | 17.5 [16.2 to 19.3] | 14.2 [12.9 to 15.5]
  Final Analysis | 18.1 [16.2 to 19.5] | 14.2 [12.9 to 15.7]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Primary Analysis. The null hypothesis is that the survival distribution of OS is the same in the two treatment arms; Test type: Superiority — The study was designed to have 80% power to show a significant difference with respect to the primary endpoint; p = 0.0565, Stratified Log-Rank — The actual p-value significance threshold required for OS was 0.0455, after alpha spent at the interim analysis was taken into account; Stratified analysis by geographic region, HER2 status, and prior gastrectomy; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 1.00] — HR was calculated as pertuzumab arm vs. placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Final Analysis; Test type: Other — Exploratory; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.72 to 0.99] — HR was calculated as pertuzumab arm vs. placebo arm. Stratified analysis by geographic region, HER2 status, and prior gastrectomy

2. Secondary Outcome: Progression-Free Survival, as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: Progression-free survival (PFS) is defined as the time from randomization to the first occurrence of progressive disease (PD), as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Tumor assessments with CT or MRI scans of the chest, abdomen, and pelvis were performed every 9 weeks. Participants without documented PD or death were censored at the tumor assessment date for which the participant was last known to be progression-free. Participants who did not have any post-baseline tumor assessment data were censored at the date of randomization plus 1 day. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 millimeters (mm) in the sum of diameters of target lesions; the appearance of one or more new lesions.
Time Frame: Baseline to death or progressive disease (PD), whichever occurred first (Median [full range] duration of follow-up in Pertuzumab vs. Placebo arms for Primary Analysis: 24.9 [0-41] vs. 21.3 [0-39] months; Final Analysis: 50.4 [0-70] vs. 47.4 [0-66] months)
Population: The ITT population included all randomized participants, regardless of whether study medication was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 388 | 392
months
  Primary Analysis | 8.5 [8.2 to 9.7] | 7.0 [6.4 to 8.2]
  Final Analysis | 8.5 [8.3 to 9.7] | 7.2 [6.4 to 8.2]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Primary Analysis; Test type: Superiority; As pre-specified in the protocol, a p-value was only to be calculated for PFS if OS was statistically significant; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.86] — A stratified Cox proportional hazards regression model was used to estimate the HR between the pertuzumab arm vs. the placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Final Analysis; Test type: Other — Exploratory; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.85] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Primary Analysis of the Percentage of Participants With Overall Objective Response, as Determined by the Investigator According to RECIST v1.1 Criteria
Description: The overall objective response rate was defined as the percentage of participants with partial response (PR) or complete response (CR) occurring on two consecutive occasions ≥4 weeks apart, as determined by the investigator using RECIST v1.1. Tumor assessments with computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest, abdomen, and pelvis were performed every 9 weeks. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR: disappearance of all target lesions. Measurable disease is defined as tumor lesions measured in at least one dimension (longest diameter in plane of measurement) with a minimum size of: 10 mm by CT or MRI scan; 10 mm caliper measurement by clinical examination; 20 mm by chest X-ray. For a malignant lymph node to be considered pathologically enlarged and measurable, it must be greater than or equal to (≥) 15 mm in short axis when assessed by CT scan.
Time Frame: Baseline up to death or progressive disease, whichever occurred first (Median [full range] duration of follow-up in Pertuzumab vs. Placebo arms for Primary Analysis: 24.9 [0-41] months vs. 21.3 [0-39] months)
Population: The subset of participants with measurable disease at baseline, according to RECIST v1.1 criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 351 | 352
Percentage of participants
  Objective Response (CR + PR) | 56.7 [51.33 to 61.95] | 48.3 [42.97 to 53.65]
  Complete Response (CR) | 5.1 [3.07 to 7.98] | 0.9 [0.18 to 2.47]
  Partial Response (PR) | 51.6 [46.20 to 56.91] | 47.4 [42.13 to 52.80]
  Stable Disease (SD) | 27.9 [23.29 to 32.93] | 33.0 [28.06 to 38.14]
  Progressive Disease (PD) | 4.8 [2.85 to 7.64] | 8.0 [5.35 to 11.29]
  Not Evaluable/Missing | 10.5 [7.53 to 14.24] | 10.8 [7.75 to 14.52]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Primary Analysis of Objective Response Rate; Test type: Other — Exploratory; Difference in Objective Response = 8.40, 95% CI 2-sided [0.89 to 15.91] — Difference in objective response was calculated as the pertuzumab arm minus placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Primary Analysis of Objective Response Rate; Test type: Other — Exploratory; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.04 to 1.89] — Odds ratio was calculated as the pertuzumab arm vs. placebo arm

4. Secondary Outcome: Final Analysis of the Percentage of Participants With Overall Objective Response, as Determined by the Investigator According to RECIST v1.1 Criteria
Description: as for outcome 3
Time Frame: Baseline up to death or progressive disease, whichever occurred first (Median [full range] duration of follow-up in Pertuzumab vs. Placebo arms for Final Analysis: 50.4 [0-70] months vs. 47.4 [0-66] months)
Population: The subset of participants with measurable disease at baseline, according to RECIST v1.1 criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 351 | 352
Percentage of participants
  Objective Response (CR + PR) | 57.0 [51.62 to 62.22] | 48.6 [43.25 to 53.94]
  Complete Response (CR) | 5.7 [3.51 to 8.66] | 2.0 [0.80 to 4.05]
  Partial Response (PR) | 51.3 [45.92 to 56.62] | 46.6 [41.29 to 51.95]
  Stable Disease (SD) | 27.6 [23.02 to 32.63] | 32.7 [27.79 to 37.84]
  Progressive Disease (PD) | 4.8 [2.85 to 7.64] | 8.2 [5.59 to 11.62]
  Not Evaluable/Missing | 10.5 [7.53 to 14.24] | 10.5 [7.51 to 14.20]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Final Analysis of Objective Response Rate; Test type: Other — Exploratory; Difference in Objective Response = 8.40, 95% CI 2-sided [0.89 to 15.91] — Difference in objective response was calculated as the pertuzumab arm minus placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Final Analysis of Objective Response Rate; Test type: Other — Exploratory; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.04 to 1.89] — Odds ratio was calculated as the pertuzumab arm vs. placebo arm

5. Secondary Outcome: Duration of Objective Response, as Determined by Investigator According to RECIST v1.1 Criteria
Description: Duration of objective response is defined as the time from first occurrence of documented objective response to documented disease progression, as determined by the investigator using RECIST v1.1, or death from any cause. Objective response: PR or CR occurring on 2 consecutive occasions ≥4 weeks apart. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR: disappearance of all target lesions. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; the appearance of one or more new lesions. Measurable disease defined as tumor lesions with a minimum size of: 10 mm by CT or MRI scan; 10 mm caliper measurement by clinical examination; 20 mm by chest X-ray. For a malignant lymph node, it must be ≥15 mm in short axis when assessed by CT scan.
Time Frame: as for outcome 2
Population: The participants with measurable disease at baseline who achieved a documented objective response, according to RECIST v1.1 criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 200 | 171
months
  Primary Analysis: number analyzed (Participants) | 199 | 170
  Primary Analysis | 10.2 [8.4 to 10.7] | 8.4 [6.8 to 8.7]
  Final Analysis | 10.2 [8.5 to 11.6] | 8.4 [6.7 to 9.0]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Primary Analysis; Test type: Other — Exploratory; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.64 to 1.06] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Final Analysis; Test type: Other — Exploratory; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.98] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants With Clinical Benefit, as Determined by the Investigator According to RECIST v1.1 Criteria
Description: The clinical benefit rate was defined as best response of complete response (CR) or partial response (PR) or stable disease (SD) for 6 weeks or longer, as determined by the investigator using RECIST v1.1. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum diameters while on study. Measurable disease is defined as tumor lesions measured in at least one dimension (longest diameter in plane of measurement) with a minimum size of: 10 mm by CT or MRI scan; 10 mm caliper measurement by clinical examination; 20 mm by chest X-ray. For a malignant lymph node to be considered pathologically enlarged and measurable, it must be >/=15 mm in short axis when assessed by CT scan. The clinical benefit rate was not updated at the final analysis.
Time Frame: as for outcome 3
Population: The subset of participants with measurable disease at baseline, according to RECIST v1.1 criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 351 | 352
percentage of participants | 84.6 [80.41 to 88.23] | 81.3 [76.77 to 85.19]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Other — Exploratory; Difference in Clinical Benefit Rate = 3.37, 95% CI 2-sided [-2.34 to 9.07] — Difference in clinical benefit rate was calculated as the pertuzumab arm minus placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Other — Exploratory; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.86 to 1.88] — Odds ratio was calculated as the pertuzumab arm vs. placebo arm

7. Secondary Outcome: Overview of Safety: Number of Participants With at Least One Adverse Event, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. The investigator graded all AEs for severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE.
Time Frame: From Baseline until end of post-treatment follow-up (up to 70 months)
Population: The safety population included all participants who received any amount of any study medication. Those who received any amount of pertuzumab were included in the pertuzumab arm; all other treated participants were included in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 385 | 388
Participants
  Any Adverse Event (AE) | 381 | 385
  AE with Fatal Outcome | 27 | 31
  Serious AE | 178 | 156
  Grade 3-5 AE | 310 | 288
  AE Leading to Pertuz/Pbo & Trastuz Discontinuation | 48 | 46
  AE Leading to Dose Interruption &/or Dose Delay | 110 | 94

8. Secondary Outcome: Number of Participants With Symptomatic or Asymptomatic Left Ventricular Systolic Dysfunction (LVSD)
Description: The number and percentage of participants with symptomatic left ventricular systolic dysfunction (LVSD) and asymptomatic LVSD events (defined as a left ventricular ejection fraction [LVEF] ≥10% decrease from baseline to an absolute value <50%) at any time during the study was summarized by treatment arm.
Time Frame: From Baseline until end of post-treatment follow-up (up to 70 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 385 | 388
Participants
  Symptomatic LVSD | 3 | 1
  Asymptomatic LVSD | 20 | 18

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Score
Description: The EORTC QLQ-C30 included global health status, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea/vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0 - 100 scale, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be a minimally important difference to participants. A positive value means an increase, while a negative value means a decrease, in score at the indicated time-point relative to the score at baseline (Cycle 1, Day 1).
Time Frame: Day 1 of each 21-day treatment cycle up to 28 and 60-90 days (post-treatment [PT] monitoring visits 1 and 2, respectively) after Day 1 of last treatment cycle (up to approximately 3.5 years)
Population: Participants in the ITT population (includes all randomized participants, regardless of whether study medication was received) with both a baseline assessment and at least 1 post-treatment assessment are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 388 | 392
score on a scale
  Appetite Loss: Cycle 1 (Baseline): number analyzed (Participants) | 371 | 383
  Appetite Loss: Cycle 1 (Baseline) | 26.68 (28.65) | 27.59 (29.96)
  Appetite Loss: Change at Cycle 2: number analyzed (Participants) | 335 | 343
  Appetite Loss: Change at Cycle 2 | 6.57 (33.18) | 0.97 (35.86)
  Appetite Loss: Change at Cycle 3: number analyzed (Participants) | 321 | 315
  Appetite Loss: Change at Cycle 3 | 3.63 (36.19) | 3.81 (36.76)
  Appetite Loss: Change at Cycle 4: number analyzed (Participants) | 299 | 294
  Appetite Loss: Change at Cycle 4 | 5.24 (34.20) | 0.79 (34.33)
  Appetite Loss: Change at Cycle 5: number analyzed (Participants) | 286 | 287
  Appetite Loss: Change at Cycle 5 | 4.55 (36.50) | 2.90 (35.85)
  Appetite Loss: Change at Cycle 6: number analyzed (Participants) | 271 | 257
  Appetite Loss: Change at Cycle 6 | 3.94 (36.07) | -0.39 (36.86)
  Appetite Loss: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Appetite Loss: Change at Cycle 7 | 2.07 (38.05) | 1.61 (35.98)
  Appetite Loss: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Appetite Loss: Change at Cycle 8 | -2.42 (33.81) | -3.69 (34.20)
  Appetite Loss: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Appetite Loss: Change at Cycle 9 | -6.67 (31.92) | -4.76 (31.67)
  Appetite Loss: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Appetite Loss: Change at Cycle 10 | -8.06 (32.52) | -6.63 (28.48)
  Appetite Loss: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Appetite Loss: Change at Cycle 11 | -9.36 (33.19) | -9.68 (27.38)
  Appetite Loss: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Appetite Loss: Change at Cycle 12 | -9.22 (33.73) | -9.05 (28.51)
  Appetite Loss: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Appetite Loss: Change at Cycle 13 | -10.17 (31.10) | -10.81 (29.18)
  Appetite Loss: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Appetite Loss: Change at Cycle 14 | -12.10 (31.96) | -12.09 (30.32)
  Appetite Loss: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Appetite Loss: Change at Cycle 15 | -8.21 (32.96) | -9.18 (29.81)
  Appetite Loss: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Appetite Loss: Change at Cycle 16 | -6.03 (33.07) | -10.59 (28.74)
  Appetite Loss: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Appetite Loss: Change at Cycle 17 | -6.55 (29.29) | -9.91 (29.05)
  Appetite Loss: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Appetite Loss: Change at Cycle 18 | -4.90 (31.25) | -14.08 (27.98)
  Appetite Loss: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Appetite Loss: Change at Cycle 19 | -8.33 (31.34) | -13.13 (28.57)
  Appetite Loss: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Appetite Loss: Change at Cycle 20 | -3.97 (31.65) | -13.23 (29.66)
  Appetite Loss: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Appetite Loss: Change at Cycle 21 | -5.91 (31.01) | -14.20 (32.76)
  Appetite Loss: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Appetite Loss: Change at Cycle 22 | -4.98 (34.45) | -16.31 (29.38)
  Appetite Loss: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Appetite Loss: Change at Cycle 23 | -6.35 (36.84) | -11.36 (35.90)
  Appetite Loss: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Appetite Loss: Change at Cycle 24 | -7.78 (33.82) | -13.33 (30.00)
  Appetite Loss: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Appetite Loss: Change at Cycle 25 | -7.05 (35.14) | -12.04 (31.02)
  Appetite Loss: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Appetite Loss: Change at Cycle 26 | -7.48 (34.87) | -12.50 (32.52)
  Appetite Loss: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Appetite Loss: Change at Cycle 27 | -10.08 (33.76) | -9.20 (28.03)
  Appetite Loss: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Appetite Loss: Change at Cycle 28 | -10.00 (32.20) | -11.54 (29.73)
  Appetite Loss: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Appetite Loss: Change at PT Visit 1 | 7.30 (36.86) | 2.64 (33.14)
  Appetite Loss: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Appetite Loss: Change at PT Visit 2 | -0.33 (33.83) | 4.55 (34.53)
  Cognitive Functional Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 382
  Cognitive Functional Scale: Cycle 1 (Baseline) | 87.95 (17.32) | 88.22 (16.18)
  Cognitive Functional Scale: Change at Cycle 2: number analyzed (Participants) | 333 | 341
  Cognitive Functional Scale: Change at Cycle 2 | -1.90 (17.82) | -1.81 (16.93)
  Cognitive Functional Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 315
  Cognitive Functional Scale: Change at Cycle 3 | -0.83 (17.11) | -3.17 (18.30)
  Cognitive Functional Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 295
  Cognitive Functional Scale: Change at Cycle 4 | -2.04 (17.78) | -2.99 (19.28)
  Cognitive Functional Scale: Change at Cycle 5: number analyzed (Participants) | 285 | 287
  Cognitive Functional Scale: Change at Cycle 5 | -3.04 (19.09) | -4.59 (19.59)
  Cognitive Functional Scale: Change at Cycle 6: number analyzed (Participants) | 271 | 256
  Cognitive Functional Scale: Change at Cycle 6 | -5.10 (19.23) | -3.84 (19.00)
  Cognitive Functional Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Cognitive Functional Scale: Change at Cycle 7 | -4.34 (19.52) | -4.31 (19.09)
  Cognitive Functional Scale: Change at Cycle 8: number analyzed (Participants) | 233 | 217
  Cognitive Functional Scale: Change at Cycle 8 | -3.15 (17.90) | -3.30 (17.59)
  Cognitive Functional Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Cognitive Functional Scale: Change at Cycle 9 | -2.22 (18.53) | -4.59 (18.53)
  Cognitive Functional Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Cognitive Functional Scale: Change at Cycle 10 | -3.32 (19.44) | -3.11 (18.50)
  Cognitive Functional Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Cognitive Functional Scale: Change at Cycle 11 | -2.83 (18.44) | -3.44 (17.06)
  Cognitive Functional Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 139
  Cognitive Functional Scale: Change at Cycle 12 | -3.35 (20.00) | -2.52 (18.16)
  Cognitive Functional Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Cognitive Functional Scale: Change at Cycle 13 | -1.79 (19.04) | -3.60 (17.89)
  Cognitive Functional Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Cognitive Functional Scale: Change at Cycle 14 | -1.98 (19.00) | -2.29 (17.56)
  Cognitive Functional Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Cognitive Functional Scale: Change at Cycle 15 | -1.15 (18.47) | -2.38 (16.05)
  Cognitive Functional Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Cognitive Functional Scale: Change at Cycle 16 | -2.73 (17.16) | -2.55 (17.16)
  Cognitive Functional Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Cognitive Functional Scale: Change at Cycle 17 | -2.53 (17.21) | -1.13 (15.44)
  Cognitive Functional Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Cognitive Functional Scale: Change at Cycle 18 | -2.78 (18.18) | 0.47 (16.42)
  Cognitive Functional Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Cognitive Functional Scale: Change at Cycle 19 | -1.04 (18.07) | 0.00 (14.62)
  Cognitive Functional Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Cognitive Functional Scale: Change at Cycle 20 | -2.18 (19.67) | 0.79 (15.68)
  Cognitive Functional Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Cognitive Functional Scale: Change at Cycle 21 | -2.11 (20.56) | 0.62 (16.50)
  Cognitive Functional Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Cognitive Functional Scale: Change at Cycle 22 | -4.73 (18.98) | -0.71 (18.04)
  Cognitive Functional Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Cognitive Functional Scale: Change at Cycle 23 | -2.38 (19.60) | 1.14 (17.75)
  Cognitive Functional Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Cognitive Functional Scale: Change at Cycle 24 | -2.78 (19.69) | 1.25 (16.18)
  Cognitive Functional Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Cognitive Functional Scale: Change at Cycle 25 | -5.45 (16.41) | -0.93 (18.66)
  Cognitive Functional Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Cognitive Functional Scale: Change at Cycle 26 | -2.38 (16.32) | -1.56 (18.63)
  Cognitive Functional Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Cognitive Functional Scale: Change at Cycle 27 | -3.88 (18.84) | -1.15 (18.33)
  Cognitive Functional Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Cognitive Functional Scale: Change at Cycle 28 | -3.75 (15.78) | 0.00 (20.00)
  Cognitive Functional Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Cognitive Functional Scale: Change at PT Visit 1 | -9.13 (21.90) | -9.16 (20.02)
  Cognitive Functional Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Cognitive Functional Scale: Change at PT Visit 2 | -8.42 (20.22) | -11.21 (22.48)
  Constipation Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 382
  Constipation Symptom Scale: Cycle 1 (Baseline) | 20.43 (28.45) | 18.41 (27.13)
  Constipation Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 334 | 341
  Constipation Symptom Scale: Change at Cycle 2 | -5.39 (27.05) | 0.29 (27.23)
  Constipation Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 316
  Constipation Symptom Scale: Change at Cycle 3 | -7.48 (28.98) | -2.11 (27.65)
  Constipation Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 295
  Constipation Symptom Scale: Change at Cycle 4 | -5.32 (29.21) | -3.73 (28.26)
  Constipation Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 287
  Constipation Symptom Scale: Change at Cycle 5 | -5.94 (29.15) | -1.28 (27.64)
  Constipation Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 271 | 257
  Constipation Symptom Scale: Change at Cycle 6 | -7.13 (29.65) | -2.33 (30.24)
  Constipation Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Constipation Symptom Scale: Change at Cycle 7 | -8.13 (30.11) | -4.09 (29.06)
  Constipation Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 232 | 217
  Constipation Symptom Scale: Change at Cycle 8 | -8.05 (30.90) | -4.45 (27.32)
  Constipation Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Constipation Symptom Scale: Change at Cycle 9 | -10.00 (27.10) | -5.61 (26.74)
  Constipation Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Constipation Symptom Scale: Change at Cycle 10 | -9.32 (29.56) | -7.43 (26.81)
  Constipation Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Constipation Symptom Scale: Change at Cycle 11 | -9.16 (29.60) | -6.88 (27.84)
  Constipation Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Constipation Symptom Scale: Change at Cycle 12 | -10.27 (29.04) | -7.25 (25.39)
  Constipation Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 110
  Constipation Symptom Scale: Change at Cycle 13 | -11.19 (29.55) | -5.76 (26.27)
  Constipation Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Constipation Symptom Scale: Change at Cycle 14 | -11.60 (27.11) | -6.21 (26.00)
  Constipation Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Constipation Symptom Scale: Change at Cycle 15 | -10.51 (26.59) | -7.14 (24.52)
  Constipation Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Constipation Symptom Scale: Change at Cycle 16 | -8.62 (24.91) | -7.45 (25.39)
  Constipation Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Constipation Symptom Scale: Change at Cycle 17 | -8.33 (24.30) | -5.86 (18.59)
  Constipation Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Constipation Symptom Scale: Change at Cycle 18 | -7.52 (22.93) | -6.57 (26.20)
  Constipation Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Constipation Symptom Scale: Change at Cycle 19 | -3.47 (25.81) | -3.03 (25.97)
  Constipation Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Constipation Symptom Scale: Change at Cycle 20 | -3.97 (26.08) | -4.76 (26.68)
  Constipation Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Constipation Symptom Scale: Change at Cycle 21 | -3.80 (29.23) | -9.26 (25.42)
  Constipation Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Constipation Symptom Scale: Change at Cycle 22 | -4.98 (28.58) | -8.51 (27.34)
  Constipation Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Constipation Symptom Scale: Change at Cycle 23 | -6.35 (28.62) | -8.33 (26.04)
  Constipation Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Constipation Symptom Scale: Change at Cycle 24 | -7.78 (27.01) | -10.00 (26.37)
  Constipation Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Constipation Symptom Scale: Change at Cycle 25 | -7.05 (29.77) | -9.26 (28.30)
  Constipation Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Constipation Symptom Scale: Change at Cycle 26 | -6.12 (30.94) | -6.25 (23.09)
  Constipation Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Constipation Symptom Scale: Change at Cycle 27 | -7.75 (28.95) | -10.34 (26.88)
  Constipation Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Constipation Symptom Scale: Change at Cycle 28 | -6.67 (26.37) | -6.41 (21.12)
  Constipation Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Constipation Symptom Scale: Change at PT Visit 1 | -6.78 (31.45) | -4.62 (26.19)
  Constipation Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Constipation Symptom Scale: Change at PT Visit 2 | -6.93 (28.41) | -0.91 (31.11)
  Diarrhea Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 382
  Diarrhea Symptom Scale: Cycle 1 (Baseline) | 8.87 (17.70) | 9.16 (18.87)
  Diarrhea Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 333 | 340
  Diarrhea Symptom Scale: Change at Cycle 2 | 15.12 (30.42) | 5.20 (23.79)
  Diarrhea Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 314
  Diarrhea Symptom Scale: Change at Cycle 3 | 14.64 (27.71) | 4.99 (26.10)
  Diarrhea Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 295
  Diarrhea Symptom Scale: Change at Cycle 4 | 14.13 (27.15) | 4.63 (24.07)
  Diarrhea Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 287
  Diarrhea Symptom Scale: Change at Cycle 5 | 13.17 (25.47) | 4.99 (23.70)
  Diarrhea Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 270 | 256
  Diarrhea Symptom Scale: Change at Cycle 6 | 14.81 (27.01) | 2.47 (23.76)
  Diarrhea Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Diarrhea Symptom Scale: Change at Cycle 7 | 12.26 (23.74) | 2.92 (23.44)
  Diarrhea Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 232 | 217
  Diarrhea Symptom Scale: Change at Cycle 8 | 8.91 (23.56) | 2.61 (23.53)
  Diarrhea Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Diarrhea Symptom Scale: Change at Cycle 9 | 6.83 (23.76) | 2.04 (21.25)
  Diarrhea Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Diarrhea Symptom Scale: Change at Cycle 10 | 6.63 (23.97) | 0.60 (20.91)
  Diarrhea Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 154
  Diarrhea Symptom Scale: Change at Cycle 11 | 5.26 (21.80) | 2.60 (20.36)
  Diarrhea Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 139
  Diarrhea Symptom Scale: Change at Cycle 12 | 3.98 (22.30) | 1.92 (19.97)
  Diarrhea Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Diarrhea Symptom Scale: Change at Cycle 13 | 4.29 (24.27) | 1.50 (19.27)
  Diarrhea Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Diarrhea Symptom Scale: Change at Cycle 14 | 3.95 (24.45) | 0.98 (20.15)
  Diarrhea Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Diarrhea Symptom Scale: Change at Cycle 15 | 3.33 (23.79) | 1.02 (19.42)
  Diarrhea Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Diarrhea Symptom Scale: Change at Cycle 16 | 5.46 (21.06) | 3.14 (15.10)
  Diarrhea Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Diarrhea Symptom Scale: Change at Cycle 17 | 2.68 (21.05) | 2.25 (14.94)
  Diarrhea Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Diarrhea Symptom Scale: Change at Cycle 18 | 3.59 (21.95) | 3.29 (17.95)
  Diarrhea Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Diarrhea Symptom Scale: Change at Cycle 19 | 3.82 (19.86) | 2.02 (16.41)
  Diarrhea Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Diarrhea Symptom Scale: Change at Cycle 20 | 5.95 (19.47) | 3.70 (17.05)
  Diarrhea Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Diarrhea Symptom Scale: Change at Cycle 21 | 3.80 (23.26) | 1.85 (16.40)
  Diarrhea Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Diarrhea Symptom Scale: Change at Cycle 22 | 6.97 (24.98) | 4.26 (17.88)
  Diarrhea Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Diarrhea Symptom Scale: Change at Cycle 23 | 6.88 (21.72) | 8.33 (20.49)
  Diarrhea Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Diarrhea Symptom Scale: Change at Cycle 24 | 7.22 (22.21) | 3.33 (16.54)
  Diarrhea Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Diarrhea Symptom Scale: Change at Cycle 25 | 8.97 (23.91) | 2.78 (14.64)
  Diarrhea Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Diarrhea Symptom Scale: Change at Cycle 26 | 5.44 (21.89) | 5.21 (20.93)
  Diarrhea Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Diarrhea Symptom Scale: Change at Cycle 27 | 3.88 (22.07) | 3.45 (16.29)
  Diarrhea Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Diarrhea Symptom Scale: Change at Cycle 28 | 7.50 (27.72) | 2.56 (16.12)
  Diarrhea Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 176 | 202
  Diarrhea Symptom Scale: Change at PT Visit 1 | 8.14 (26.00) | 1.98 (24.35)
  Diarrhea Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Diarrhea Symptom Scale: Change at PT Visit 2 | 7.26 (25.65) | 4.24 (29.65)
  Dyspnoea Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 370 | 382
  Dyspnoea Symptom Scale: Cycle 1 (Baseline) | 12.07 (17.99) | 12.65 (20.20)
  Dyspnoea Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 335 | 341
  Dyspnoea Symptom Scale: Change at Cycle 2 | -0.50 (19.04) | 0.29 (19.72)
  Dyspnoea Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 320 | 314
  Dyspnoea Symptom Scale: Change at Cycle 3 | -0.31 (20.18) | -0.32 (20.38)
  Dyspnoea Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 299 | 294
  Dyspnoea Symptom Scale: Change at Cycle 4 | 1.23 (20.31) | 1.81 (21.08)
  Dyspnoea Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 284 | 287
  Dyspnoea Symptom Scale: Change at Cycle 5 | 2.58 (20.62) | 1.39 (21.18)
  Dyspnoea Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 271 | 256
  Dyspnoea Symptom Scale: Change at Cycle 6 | 3.20 (23.79) | 0.39 (20.55)
  Dyspnoea Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 241 | 227
  Dyspnoea Symptom Scale: Change at Cycle 7 | 0.00 (21.94) | 0.59 (20.07)
  Dyspnoea Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 233 | 216
  Dyspnoea Symptom Scale: Change at Cycle 8 | -0.14 (21.99) | 0.93 (20.56)
  Dyspnoea Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 209 | 196
  Dyspnoea Symptom Scale: Change at Cycle 9 | -1.12 (20.51) | 0.17 (18.95)
  Dyspnoea Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 185 | 166
  Dyspnoea Symptom Scale: Change at Cycle 10 | -0.54 (21.56) | 1.00 (16.99)
  Dyspnoea Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 170 | 155
  Dyspnoea Symptom Scale: Change at Cycle 11 | -2.16 (19.58) | -1.29 (17.77)
  Dyspnoea Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 158 | 140
  Dyspnoea Symptom Scale: Change at Cycle 12 | -2.53 (19.75) | -0.71 (18.95)
  Dyspnoea Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Dyspnoea Symptom Scale: Change at Cycle 13 | -1.43 (20.34) | -1.20 (16.77)
  Dyspnoea Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Dyspnoea Symptom Scale: Change at Cycle 14 | -1.98 (19.00) | -2.61 (17.98)
  Dyspnoea Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 129 | 98
  Dyspnoea Symptom Scale: Change at Cycle 15 | -2.84 (21.26) | 2.72 (18.95)
  Dyspnoea Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 115 | 85
  Dyspnoea Symptom Scale: Change at Cycle 16 | -1.45 (20.42) | 1.18 (18.86)
  Dyspnoea Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 110 | 74
  Dyspnoea Symptom Scale: Change at Cycle 17 | -1.82 (20.61) | 0.90 (19.87)
  Dyspnoea Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Dyspnoea Symptom Scale: Change at Cycle 18 | -0.98 (20.15) | -2.35 (18.10)
  Dyspnoea Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Dyspnoea Symptom Scale: Change at Cycle 19 | -1.74 (20.73) | 0.51 (18.15)
  Dyspnoea Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Dyspnoea Symptom Scale: Change at Cycle 20 | -1.19 (20.98) | -1.06 (16.90)
  Dyspnoea Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Dyspnoea Symptom Scale: Change at Cycle 21 | 1.27 (22.29) | -0.62 (19.95)
  Dyspnoea Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Dyspnoea Symptom Scale: Change at Cycle 22 | -1.99 (22.38) | 0.71 (14.73)
  Dyspnoea Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Dyspnoea Symptom Scale: Change at Cycle 23 | -1.59 (21.94) | 1.52 (14.30)
  Dyspnoea Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Dyspnoea Symptom Scale: Change at Cycle 24 | 1.11 (22.10) | -1.67 (12.96)
  Dyspnoea Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Dyspnoea Symptom Scale: Change at Cycle 25 | 0.64 (21.38) | -3.70 (15.49)
  Dyspnoea Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Dyspnoea Symptom Scale: Change at Cycle 26 | 0.00 (22.57) | 1.04 (23.16)
  Dyspnoea Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Dyspnoea Symptom Scale: Change at Cycle 27 | 0.78 (21.19) | 3.45 (22.44)
  Dyspnoea Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Dyspnoea Symptom Scale: Change at Cycle 28 | 1.67 (21.28) | 3.85 (17.20)
  Dyspnoea Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Dyspnoea Symptom Scale: Change at PT Visit 1 | 6.97 (26.98) | 6.77 (23.82)
  Dyspnoea Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Dyspnoea Symptom Scale: Change at PT Visit 2 | 3.30 (23.81) | 9.39 (26.76)
  Emotional Functional Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 382
  Emotional Functional Scale: Cycle 1 (Baseline) | 76.90 (20.21) | 76.56 (19.84)
  Emotional Functional Scale: Change at Cycle 2: number analyzed (Participants) | 333 | 341
  Emotional Functional Scale: Change at Cycle 2 | 3.53 (16.84) | 3.05 (18.49)
  Emotional Functional Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 315
  Emotional Functional Scale: Change at Cycle 3 | 2.65 (18.63) | 3.96 (19.95)
  Emotional Functional Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 295
  Emotional Functional Scale: Change at Cycle 4 | 3.10 (21.11) | 3.67 (20.44)
  Emotional Functional Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 287
  Emotional Functional Scale: Change at Cycle 5 | 2.62 (19.97) | 2.74 (21.72)
  Emotional Functional Scale: Change at Cycle 6: number analyzed (Participants) | 271 | 256
  Emotional Functional Scale: Change at Cycle 6 | 1.01 (19.64) | 4.93 (21.00)
  Emotional Functional Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Emotional Functional Scale: Change at Cycle 7 | 1.72 (21.09) | 4.41 (20.18)
  Emotional Functional Scale: Change at Cycle 8: number analyzed (Participants) | 233 | 217
  Emotional Functional Scale: Change at Cycle 8 | 3.43 (20.66) | 5.66 (19.63)
  Emotional Functional Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Emotional Functional Scale: Change at Cycle 9 | 4.72 (20.10) | 4.78 (19.45)
  Emotional Functional Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Emotional Functional Scale: Change at Cycle 10 | 3.72 (21.76) | 6.74 (18.13)
  Emotional Functional Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Emotional Functional Scale: Change at Cycle 11 | 5.85 (19.64) | 4.96 (19.21)
  Emotional Functional Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 139
  Emotional Functional Scale: Change at Cycle 12 | 4.93 (21.38) | 5.24 (19.14)
  Emotional Functional Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Emotional Functional Scale: Change at Cycle 13 | 5.00 (23.07) | 5.18 (17.95)
  Emotional Functional Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Emotional Functional Scale: Change at Cycle 14 | 5.93 (22.90) | 6.29 (19.03)
  Emotional Functional Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Emotional Functional Scale: Change at Cycle 15 | 6.03 (22.13) | 5.19 (19.61)
  Emotional Functional Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Emotional Functional Scale: Change at Cycle 16 | 5.17 (23.20) | 5.29 (20.81)
  Emotional Functional Scale: Change at Cycle 17: number analyzed (Participants) | 111 | 74
  Emotional Functional Scale: Change at Cycle 17 | 6.01 (23.55) | 6.31 (18.70)
  Emotional Functional Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Emotional Functional Scale: Change at Cycle 18 | 3.68 (24.11) | 5.87 (19.39)
  Emotional Functional Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Emotional Functional Scale: Change at Cycle 19 | 4.69 (26.01) | 5.56 (18.68)
  Emotional Functional Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Emotional Functional Scale: Change at Cycle 20 | 3.47 (26.92) | 5.42 (17.91)
  Emotional Functional Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Emotional Functional Scale: Change at Cycle 21 | 4.54 (26.55) | 6.48 (22.00)
  Emotional Functional Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Emotional Functional Scale: Change at Cycle 22 | 5.35 (28.67) | 6.91 (18.66)
  Emotional Functional Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Emotional Functional Scale: Change at Cycle 23 | 5.82 (28.42) | 6.63 (21.00)
  Emotional Functional Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Emotional Functional Scale: Change at Cycle 24 | 5.28 (26.22) | 8.54 (19.57)
  Emotional Functional Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Emotional Functional Scale: Change at Cycle 25 | 5.93 (25.48) | 8.80 (20.89)
  Emotional Functional Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Emotional Functional Scale: Change at Cycle 26 | 5.44 (27.77) | 5.99 (16.15)
  Emotional Functional Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Emotional Functional Scale: Change at Cycle 27 | 7.56 (28.34) | 5.75 (18.51)
  Emotional Functional Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Emotional Functional Scale: Change at Cycle 28 | 7.08 (25.43) | 7.05 (18.96)
  Emotional Functional Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Emotional Functional Scale: Change at PT Visit 1 | -5.48 (23.16) | -3.92 (23.28)
  Emotional Functional Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Emotional Functional Scale: Change at PT Visit 2 | -2.64 (23.33) | -4.47 (23.34)
  Fatigue Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 383
  Fatigue Symptom Scale: Cycle 1 (Baseline) | 31.96 (23.46) | 32.27 (21.92)
  Fatigue Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 336 | 343
  Fatigue Symptom Scale: Change at Cycle 2 | 3.13 (19.80) | 2.32 (21.57)
  Fatigue Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 322 | 315
  Fatigue Symptom Scale: Change at Cycle 3 | 1.41 (22.65) | 3.19 (22.97)
  Fatigue Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 295
  Fatigue Symptom Scale: Change at Cycle 4 | 2.77 (23.14) | 1.58 (24.04)
  Fatigue Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Fatigue Symptom Scale: Change at Cycle 5 | 3.87 (25.75) | 3.05 (24.29)
  Fatigue Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Fatigue Symptom Scale: Change at Cycle 6 | 4.37 (25.64) | 2.62 (23.68)
  Fatigue Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Fatigue Symptom Scale: Change at Cycle 7 | 2.36 (26.79) | 0.97 (23.44)
  Fatigue Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Fatigue Symptom Scale: Change at Cycle 8 | -0.19 (25.00) | -1.18 (22.74)
  Fatigue Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Fatigue Symptom Scale: Change at Cycle 9 | -2.38 (22.69) | -2.01 (22.84)
  Fatigue Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Fatigue Symptom Scale: Change at Cycle 10 | -3.41 (24.69) | -3.08 (22.41)
  Fatigue Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Fatigue Symptom Scale: Change at Cycle 11 | -4.35 (22.66) | -3.44 (21.21)
  Fatigue Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Fatigue Symptom Scale: Change at Cycle 12 | -3.14 (24.56) | -4.60 (24.39)
  Fatigue Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Fatigue Symptom Scale: Change at Cycle 13 | -4.57 (23.31) | -4.50 (21.47)
  Fatigue Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Fatigue Symptom Scale: Change at Cycle 14 | -6.75 (24.32) | -6.54 (22.89)
  Fatigue Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Fatigue Symptom Scale: Change at Cycle 15 | -5.47 (24.68) | -4.99 (22.40)
  Fatigue Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Fatigue Symptom Scale: Change at Cycle 16 | -3.54 (24.81) | -6.93 (21.89)
  Fatigue Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Fatigue Symptom Scale: Change at Cycle 17 | -4.27 (25.50) | -3.45 (21.91)
  Fatigue Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Fatigue Symptom Scale: Change at Cycle 18 | -4.14 (24.42) | -8.92 (20.54)
  Fatigue Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Fatigue Symptom Scale: Change at Cycle 19 | -5.32 (27.83) | -9.01 (20.71)
  Fatigue Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Fatigue Symptom Scale: Change at Cycle 20 | -5.56 (26.64) | -6.53 (21.83)
  Fatigue Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Fatigue Symptom Scale: Change at Cycle 21 | -3.94 (25.97) | -7.41 (23.45)
  Fatigue Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Fatigue Symptom Scale: Change at Cycle 22 | -1.49 (25.58) | -10.64 (22.22)
  Fatigue Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Fatigue Symptom Scale: Change at Cycle 23 | -5.82 (25.23) | -9.60 (28.01)
  Fatigue Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Fatigue Symptom Scale: Change at Cycle 24 | -1.67 (27.05) | -12.50 (24.29)
  Fatigue Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Fatigue Symptom Scale: Change at Cycle 25 | -4.70 (26.16) | -12.35 (22.03)
  Fatigue Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Fatigue Symptom Scale: Change at Cycle 26 | -4.99 (24.85) | -11.46 (22.84)
  Fatigue Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Fatigue Symptom Scale: Change at Cycle 27 | -6.98 (23.76) | -5.36 (23.87)
  Fatigue Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Fatigue Symptom Scale: Change at Cycle 28 | -6.39 (18.98) | -4.70 (26.14)
  Fatigue Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Fatigue Symptom Scale: Change at PT Visit 1 | 10.02 (28.48) | 5.25 (24.00)
  Fatigue Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Fatigue Symptom Scale: Change at PT Visit 2 | 7.70 (27.65) | 9.70 (25.01)
  Financial Difficulties Scale: Cycle 1 (Baseline): number analyzed (Participants) | 370 | 379
  Financial Difficulties Scale: Cycle 1 (Baseline) | 26.67 (30.32) | 26.21 (29.78)
  Financial Difficulties Scale: Change at Cycle 2: number analyzed (Participants) | 332 | 339
  Financial Difficulties Scale: Change at Cycle 2 | -0.90 (26.85) | -2.46 (25.46)
  Financial Difficulties Scale: Change at Cycle 3: number analyzed (Participants) | 320 | 312
  Financial Difficulties Scale: Change at Cycle 3 | 0.31 (27.62) | 0.00 (26.33)
  Financial Difficulties Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 292
  Financial Difficulties Scale: Change at Cycle 4 | 0.89 (25.95) | 0.11 (25.10)
  Financial Difficulties Scale: Change at Cycle 5: number analyzed (Participants) | 285 | 284
  Financial Difficulties Scale: Change at Cycle 5 | 1.75 (27.71) | 2.58 (26.46)
  Financial Difficulties Scale: Change at Cycle 6: number analyzed (Participants) | 270 | 255
  Financial Difficulties Scale: Change at Cycle 6 | 1.11 (27.62) | 0.92 (26.36)
  Financial Difficulties Scale: Change at Cycle 7: number analyzed (Participants) | 240 | 224
  Financial Difficulties Scale: Change at Cycle 7 | 1.11 (31.08) | 0.30 (26.41)
  Financial Difficulties Scale: Change at Cycle 8: number analyzed (Participants) | 232 | 215
  Financial Difficulties Scale: Change at Cycle 8 | 1.15 (30.21) | 0.47 (25.27)
  Financial Difficulties Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 195
  Financial Difficulties Scale: Change at Cycle 9 | 1.11 (29.78) | -0.51 (24.75)
  Financial Difficulties Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 165
  Financial Difficulties Scale: Change at Cycle 10 | 0.90 (30.10) | -2.42 (24.30)
  Financial Difficulties Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 154
  Financial Difficulties Scale: Change at Cycle 11 | 0.39 (29.37) | -0.22 (24.84)
  Financial Difficulties Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Financial Difficulties Scale: Change at Cycle 12 | -1.05 (28.91) | -0.97 (26.39)
  Financial Difficulties Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Financial Difficulties Scale: Change at Cycle 13 | -0.95 (28.82) | 0.30 (24.82)
  Financial Difficulties Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Financial Difficulties Scale: Change at Cycle 14 | -1.73 (29.74) | -0.98 (25.02)
  Financial Difficulties Scale: Change at Cycle 15: number analyzed (Participants) | 129 | 98
  Financial Difficulties Scale: Change at Cycle 15 | -1.81 (28.96) | 1.36 (26.18)
  Financial Difficulties Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Financial Difficulties Scale: Change at Cycle 16 | -3.16 (30.13) | 0.39 (25.97)
  Financial Difficulties Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Financial Difficulties Scale: Change at Cycle 17 | -3.87 (29.59) | 1.35 (27.28)
  Financial Difficulties Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Financial Difficulties Scale: Change at Cycle 18 | -2.29 (27.46) | 2.35 (26.02)
  Financial Difficulties Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Financial Difficulties Scale: Change at Cycle 19 | -0.35 (28.41) | -0.51 (27.73)
  Financial Difficulties Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Financial Difficulties Scale: Change at Cycle 20 | 1.19 (29.47) | 1.59 (27.71)
  Financial Difficulties Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Financial Difficulties Scale: Change at Cycle 21 | 1.27 (28.96) | -4.94 (27.78)
  Financial Difficulties Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Financial Difficulties Scale: Change at Cycle 22 | 2.49 (26.79) | -4.26 (23.69)
  Financial Difficulties Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Financial Difficulties Scale: Change at Cycle 23 | -0.53 (26.43) | -2.27 (29.11)
  Financial Difficulties Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Financial Difficulties Scale: Change at Cycle 24 | 1.11 (24.52) | -5.83 (26.03)
  Financial Difficulties Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Financial Difficulties Scale: Change at Cycle 25 | 3.21 (27.42) | -4.63 (25.39)
  Financial Difficulties Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 30
  Financial Difficulties Scale: Change at Cycle 26 | 2.72 (28.74) | -2.22 (26.16)
  Financial Difficulties Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Financial Difficulties Scale: Change at Cycle 27 | -3.10 (23.92) | 1.15 (24.37)
  Financial Difficulties Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Financial Difficulties Scale: Change at Cycle 28 | -1.67 (23.81) | -1.28 (24.00)
  Financial Difficulties Scale: Change at PT Visit 1: number analyzed (Participants) | 176 | 201
  Financial Difficulties Scale: Change at PT Visit 1 | 1.70 (29.66) | 1.33 (26.21)
  Financial Difficulties Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Financial Difficulties Scale: Change at PT Visit 2 | 1.98 (26.17) | 4.24 (31.32)
  Nausea and Vomiting Scale: Cycle 1 (Baseline): number analyzed (Participants) | 371 | 383
  Nausea and Vomiting Scale: Cycle 1 (Baseline) | 11.14 (19.11) | 11.92 (18.76)
  Nausea And Vomiting Scale: Change at Cycle 2: number analyzed (Participants) | 336 | 343
  Nausea And Vomiting Scale: Change at Cycle 2 | 5.85 (22.65) | 4.08 (22.25)
  Nausea And Vomiting Scale: Change at Cycle 3: number analyzed (Participants) | 322 | 316
  Nausea And Vomiting Scale: Change at Cycle 3 | 5.12 (23.62) | 5.06 (21.14)
  Nausea And Vomiting Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 295
  Nausea And Vomiting Scale: Change at Cycle 4 | 4.10 (21.85) | 3.56 (23.76)
  Nausea And Vomiting Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Nausea And Vomiting Scale: Change at Cycle 5 | 5.13 (22.58) | 5.15 (23.81)
  Nausea And Vomiting Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Nausea And Vomiting Scale: Change at Cycle 6 | 4.11 (23.36) | 2.59 (21.24)
  Nausea And Vomiting Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Nausea And Vomiting Scale: Change at Cycle 7 | 2.07 (23.58) | 2.49 (22.31)
  Nausea And Vomiting Scale: Change at Cycle 8: number analyzed (Participants) | 233 | 217
  Nausea And Vomiting Scale: Change at Cycle 8 | -0.86 (20.80) | -0.77 (20.21)
  Nausea And Vomiting Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Nausea And Vomiting Scale: Change at Cycle 9 | -2.54 (20.85) | -2.98 (19.78)
  Nausea And Vomiting Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Nausea And Vomiting Scale: Change at Cycle 10 | -4.30 (18.81) | -2.81 (20.57)
  Nausea And Vomiting Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Nausea And Vomiting Scale: Change at Cycle 11 | -3.51 (18.01) | -3.66 (20.04)
  Nausea And Vomiting Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Nausea And Vomiting Scale: Change at Cycle 12 | -3.04 (18.07) | -3.45 (20.34)
  Nausea And Vomiting Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Nausea And Vomiting Scale: Change at Cycle 13 | -4.02 (16.29) | -3.60 (19.25)
  Nausea And Vomiting Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Nausea And Vomiting Scale: Change at Cycle 14 | -3.46 (19.54) | -5.72 (18.54)
  Nausea And Vomiting Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Nausea And Vomiting Scale: Change at Cycle 15 | -3.59 (16.34) | -3.91 (16.55)
  Nausea And Vomiting Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Nausea And Vomiting Scale: Change at Cycle 16 | -0.43 (20.32) | -2.55 (20.00)
  Nausea And Vomiting Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Nausea And Vomiting Scale: Change at Cycle 17 | -0.60 (17.46) | -3.15 (16.48)
  Nausea And Vomiting Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Nausea And Vomiting Scale: Change at Cycle 18 | -0.65 (16.90) | -3.52 (18.24)
  Nausea And Vomiting Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Nausea And Vomiting Scale: Change at Cycle 19 | -0.87 (18.32) | -4.04 (19.62)
  Nausea And Vomiting Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Nausea And Vomiting Scale: Change at Cycle 20 | -1.79 (18.48) | -3.97 (17.89)
  Nausea And Vomiting Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Nausea And Vomiting Scale: Change at Cycle 21 | -1.05 (20.03) | -6.48 (19.80)
  Nausea And Vomiting Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Nausea And Vomiting Scale: Change at Cycle 22 | -3.48 (19.14) | -8.16 (18.99)
  Nausea And Vomiting Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Nausea And Vomiting Scale: Change at Cycle 23 | -4.23 (17.70) | -6.44 (24.70)
  Nausea And Vomiting Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Nausea And Vomiting Scale: Change at Cycle 24 | -4.72 (16.26) | -7.92 (17.70)
  Nausea And Vomiting Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Nausea And Vomiting Scale: Change at Cycle 25 | -4.17 (20.84) | -7.41 (19.29)
  Nausea And Vomiting Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Nausea And Vomiting Scale: Change at Cycle 26 | -3.40 (24.29) | -9.38 (19.37)
  Nausea And Vomiting Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Nausea And Vomiting Scale: Change at Cycle 27 | -5.04 (22.58) | -7.47 (20.70)
  Nausea And Vomiting Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Nausea And Vomiting Scale: Change at Cycle 28 | -1.25 (20.11) | -6.41 (17.69)
  Nausea and Vomiting Scale: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Nausea and Vomiting Scale: Change at PT Visit 1 | 4.68 (22.20) | 4.13 (23.91)
  Nausea and Vomiting Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Nausea and Vomiting Scale: Change at PT Visit 2 | 4.29 (23.05) | 2.73 (21.60)
  Pain Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 383
  Pain Symptom Scale: Cycle 1 (Baseline) | 23.92 (25.92) | 23.72 (24.82)
  Pain Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 336 | 342
  Pain Symptom Scale: Change at Cycle 2 | -6.80 (24.69) | -6.38 (23.58)
  Pain Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 322 | 316
  Pain Symptom Scale: Change at Cycle 3 | -9.89 (25.16) | -7.23 (25.78)
  Pain Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 295
  Pain Symptom Scale: Change at Cycle 4 | -10.26 (24.78) | -7.46 (26.06)
  Pain Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Pain Symptom Scale: Change at Cycle 5 | -8.86 (25.88) | -6.25 (25.42)
  Pain Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Pain Symptom Scale: Change at Cycle 6 | -8.95 (25.73) | -7.33 (24.85)
  Pain Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Pain Symptom Scale: Change at Cycle 7 | -10.95 (26.13) | -7.46 (24.79)
  Pain Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Pain Symptom Scale: Change at Cycle 8 | -9.97 (25.80) | -8.53 (22.86)
  Pain Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Pain Symptom Scale: Change at Cycle 9 | -9.29 (24.83) | -7.82 (22.98)
  Pain Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Pain Symptom Scale: Change at Cycle 10 | -9.41 (26.10) | -8.13 (22.75)
  Pain Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Pain Symptom Scale: Change at Cycle 11 | -10.33 (25.77) | -6.34 (22.97)
  Pain Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Pain Symptom Scale: Change at Cycle 12 | -10.27 (23.10) | -5.24 (25.29)
  Pain Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Pain Symptom Scale: Change at Cycle 13 | -10.28 (25.79) | -4.80 (20.27)
  Pain Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Pain Symptom Scale: Change at Cycle 14 | -10.49 (25.49) | -5.56 (23.37)
  Pain Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Pain Symptom Scale: Change at Cycle 15 | -11.15 (22.86) | -3.74 (22.77)
  Pain Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Pain Symptom Scale: Change at Cycle 16 | -9.91 (22.94) | -4.71 (23.66)
  Pain Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Pain Symptom Scale: Change at Cycle 17 | -7.59 (25.00) | -5.63 (22.63)
  Pain Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Pain Symptom Scale: Change at Cycle 18 | -8.82 (23.42) | -8.22 (20.68)
  Pain Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Pain Symptom Scale: Change at Cycle 19 | -8.16 (25.13) | -5.05 (21.48)
  Pain Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Pain Symptom Scale: Change at Cycle 20 | -6.94 (25.90) | -6.08 (19.24)
  Pain Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Pain Symptom Scale: Change at Cycle 21 | -9.92 (27.15) | -6.48 (23.44)
  Pain Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Pain Symptom Scale: Change at Cycle 22 | -7.71 (26.96) | -8.51 (19.62)
  Pain Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Pain Symptom Scale: Change at Cycle 23 | -10.85 (22.03) | -7.95 (26.29)
  Pain Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Pain Symptom Scale: Change at Cycle 24 | -10.00 (24.39) | -10.00 (17.21)
  Pain Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Pain Symptom Scale: Change at Cycle 25 | -9.94 (24.09) | -12.96 (19.96)
  Pain Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Pain Symptom Scale: Change at Cycle 26 | -10.54 (22.49) | -8.33 (18.45)
  Pain Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Pain Symptom Scale: Change at Cycle 27 | -11.24 (22.34) | -5.75 (21.95)
  Pain Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Pain Symptom Scale: Change at Cycle 28 | -10.42 (27.91) | -9.62 (19.54)
  Pain Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Pain Symptom Scale: Change at PT Visit 1 | 1.13 (27.27) | 2.06 (28.70)
  Pain Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Pain Symptom Scale: Change at PT Visit 2 | -1.49 (28.39) | 5.45 (29.96)
  Physical Functional Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 383
  Physical Functional Scale: Cycle 1 (Baseline) | 80.86 (19.53) | 82.05 (18.32)
  Physical Functional Scale: Change at Cycle 2: number analyzed (Participants) | 336 | 343
  Physical Functional Scale: Change at Cycle 2 | -3.58 (14.56) | -3.01 (15.34)
  Physical Functional Scale: Change at Cycle 3: number analyzed (Participants) | 322 | 316
  Physical Functional Scale: Change at Cycle 3 | -2.99 (17.19) | -3.92 (17.03)
  Physical Functional Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 294
  Physical Functional Scale: Change at Cycle 4 | -3.28 (18.87) | -3.50 (17.99)
  Physical Functional Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Physical Functional Scale: Change at Cycle 5 | -3.10 (19.35) | -4.62 (17.62)
  Physical Functional Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Physical Functional Scale: Change at Cycle 6 | -5.00 (20.30) | -3.84 (18.65)
  Physical Functional Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Physical Functional Scale: Change at Cycle 7 | -3.66 (20.75) | -3.79 (19.82)
  Physical Functional Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Physical Functional Scale: Change at Cycle 8 | -2.24 (21.14) | -1.56 (18.55)
  Physical Functional Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Physical Functional Scale: Change at Cycle 9 | -1.59 (20.21) | -0.75 (18.44)
  Physical Functional Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Physical Functional Scale: Change at Cycle 10 | 0.11 (19.93) | -0.27 (17.16)
  Physical Functional Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Physical Functional Scale: Change at Cycle 11 | 0.35 (19.43) | 0.27 (17.09)
  Physical Functional Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Physical Functional Scale: Change at Cycle 12 | -1.05 (20.06) | 0.89 (16.35)
  Physical Functional Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Physical Functional Scale: Change at Cycle 13 | -0.80 (20.65) | 0.27 (17.41)
  Physical Functional Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Physical Functional Scale: Change at Cycle 14 | -0.02 (20.14) | 1.70 (18.09)
  Physical Functional Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Physical Functional Scale: Change at Cycle 15 | 0.41 (18.91) | -0.95 (17.99)
  Physical Functional Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Physical Functional Scale: Change at Cycle 16 | -1.08 (19.85) | -0.08 (18.18)
  Physical Functional Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Physical Functional Scale: Change at Cycle 17 | -0.46 (19.43) | -0.81 (17.55)
  Physical Functional Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Physical Functional Scale: Change at Cycle 18 | 0.13 (19.74) | 0.75 (16.85)
  Physical Functional Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Physical Functional Scale: Change at Cycle 19 | 1.39 (19.82) | 1.31 (14.38)
  Physical Functional Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Physical Functional Scale: Change at Cycle 20 | 0.71 (21.08) | 0.85 (16.74)
  Physical Functional Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Physical Functional Scale: Change at Cycle 21 | 0.42 (22.20) | 0.25 (18.18)
  Physical Functional Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Physical Functional Scale: Change at Cycle 22 | -2.79 (21.90) | 1.42 (16.79)
  Physical Functional Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Physical Functional Scale: Change at Cycle 23 | -1.48 (21.47) | 0.61 (19.60)
  Physical Functional Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Physical Functional Scale: Change at Cycle 24 | -2.67 (22.27) | 3.00 (16.47)
  Physical Functional Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Physical Functional Scale: Change at Cycle 25 | -2.18 (20.61) | 4.81 (15.91)
  Physical Functional Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Physical Functional Scale: Change at Cycle 26 | -1.90 (20.09) | -1.88 (20.69)
  Physical Functional Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Physical Functional Scale: Change at Cycle 27 | 0.16 (18.66) | -3.68 (19.40)
  Physical Functional Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Physical Functional Scale: Change at Cycle 28 | -1.17 (17.79) | -2.82 (18.97)
  Physical Functional Scale: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Physical Functional Scale: Change at PT Visit 1 | -11.37 (23.67) | -7.51 (20.53)
  Physical Functional Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Physical Functional Scale: Change at PT Visit 2 | -11.49 (24.31) | -11.82 (20.27)
  Global Health Status Scale: Cycle 1 (Baseline): number analyzed (Participants) | 370 | 382
  Global Health Status Scale: Cycle 1 (Baseline) | 59.77 (22.88) | 59.90 (22.11)
  Global Health Status Scale: Change at Cycle 2: number analyzed (Participants) | 331 | 340
  Global Health Status Scale: Change at Cycle 2 | 1.81 (23.35) | 4.29 (23.42)
  Global Health Status Scale: Change at Cycle 3: number analyzed (Participants) | 320 | 315
  Global Health Status Scale: Change at Cycle 3 | 1.56 (25.05) | 2.86 (25.03)
  Global Health Status Scale: Change at Cycle 4: number analyzed (Participants) | 300 | 295
  Global Health Status Scale: Change at Cycle 4 | 1.39 (25.26) | 4.15 (23.79)
  Global Health Status Scale: Change at Cycle 5: number analyzed (Participants) | 284 | 287
  Global Health Status Scale: Change at Cycle 5 | 1.17 (25.70) | 3.92 (23.05)
  Global Health Status Scale: Change at Cycle 6: number analyzed (Participants) | 268 | 256
  Global Health Status Scale: Change at Cycle 6 | 0.68 (27.89) | 3.61 (23.13)
  Global Health Status Scale: Change at Cycle 7: number analyzed (Participants) | 241 | 228
  Global Health Status Scale: Change at Cycle 7 | 1.83 (27.81) | 3.33 (22.77)
  Global Health Status Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Global Health Status Scale: Change at Cycle 8 | 3.06 (27.09) | 5.18 (23.18)
  Global Health Status Scale: Change at Cycle 9: number analyzed (Participants) | 209 | 196
  Global Health Status Scale: Change at Cycle 9 | 4.39 (26.25) | 4.68 (22.99)
  Global Health Status Scale: Change at Cycle 10: number analyzed (Participants) | 184 | 166
  Global Health Status Scale: Change at Cycle 10 | 4.80 (25.35) | 5.07 (22.77)
  Global Health Status Scale: Change at Cycle 11: number analyzed (Participants) | 170 | 155
  Global Health Status Scale: Change at Cycle 11 | 5.78 (26.62) | 3.82 (23.75)
  Global Health Status Scale: Change at Cycle 12: number analyzed (Participants) | 158 | 139
  Global Health Status Scale: Change at Cycle 12 | 3.11 (24.89) | 5.34 (24.47)
  Global Health Status Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Global Health Status Scale: Change at Cycle 13 | 3.51 (23.82) | 3.83 (23.78)
  Global Health Status Scale: Change at Cycle 14: number analyzed (Participants) | 134 | 102
  Global Health Status Scale: Change at Cycle 14 | 5.97 (23.09) | 4.82 (24.86)
  Global Health Status Scale: Change at Cycle 15: number analyzed (Participants) | 129 | 98
  Global Health Status Scale: Change at Cycle 15 | 4.26 (25.98) | 1.70 (24.46)
  Global Health Status Scale: Change at Cycle 16: number analyzed (Participants) | 115 | 85
  Global Health Status Scale: Change at Cycle 16 | 3.12 (25.16) | 3.04 (23.77)
  Global Health Status Scale: Change at Cycle 17: number analyzed (Participants) | 111 | 74
  Global Health Status Scale: Change at Cycle 17 | 2.93 (24.84) | 3.83 (24.84)
  Global Health Status Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Global Health Status Scale: Change at Cycle 18 | 3.02 (23.88) | 2.58 (27.08)
  Global Health Status Scale: Change at Cycle 19: number analyzed (Participants) | 95 | 65
  Global Health Status Scale: Change at Cycle 19 | 3.25 (26.39) | 3.97 (25.43)
  Global Health Status Scale: Change at Cycle 20: number analyzed (Participants) | 83 | 63
  Global Health Status Scale: Change at Cycle 20 | 5.12 (24.20) | 4.89 (25.69)
  Global Health Status Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Global Health Status Scale: Change at Cycle 21 | 5.38 (23.87) | 5.40 (24.72)
  Global Health Status Scale: Change at Cycle 22: number analyzed (Participants) | 66 | 47
  Global Health Status Scale: Change at Cycle 22 | 3.79 (22.56) | 3.19 (25.57)
  Global Health Status Scale: Change at Cycle 23: number analyzed (Participants) | 62 | 43
  Global Health Status Scale: Change at Cycle 23 | 4.03 (23.85) | 4.07 (27.18)
  Global Health Status Scale: Change at Cycle 24: number analyzed (Participants) | 59 | 40
  Global Health Status Scale: Change at Cycle 24 | 4.24 (22.66) | 2.92 (30.58)
  Global Health Status Scale: Change at Cycle 25: number analyzed (Participants) | 51 | 36
  Global Health Status Scale: Change at Cycle 25 | 3.59 (22.38) | 8.10 (25.39)
  Global Health Status Scale: Change at Cycle 26: number analyzed (Participants) | 47 | 32
  Global Health Status Scale: Change at Cycle 26 | 7.27 (24.55) | 5.47 (26.91)
  Global Health Status Scale: Change at Cycle 27: number analyzed (Participants) | 42 | 29
  Global Health Status Scale: Change at Cycle 27 | 7.54 (23.19) | 1.72 (28.38)
  Global Health Status Scale: Change at Cycle 28: number analyzed (Participants) | 39 | 26
  Global Health Status Scale: Change at Cycle 28 | 4.49 (22.69) | 4.81 (28.98)
  Global Health Status Scale: Change at PT Visit 1: number analyzed (Participants) | 176 | 201
  Global Health Status Scale: Change at PT Visit 1 | -7.24 (27.24) | -6.14 (24.97)
  Global Health Status Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Global Health Status Scale: Change at PT Visit 2 | -2.72 (27.46) | -5.68 (26.57)
  Role Functional Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 383
  Role Functional Scale: Cycle 1 (Baseline) | 77.06 (27.02) | 79.33 (25.12)
  Role Functional Scale: Change at Cycle 2: number analyzed (Participants) | 335 | 343
  Role Functional Scale: Change at Cycle 2 | -3.78 (24.99) | -2.82 (24.35)
  Role Functional Scale: Change at Cycle 3: number analyzed (Participants) | 322 | 315
  Role Functional Scale: Change at Cycle 3 | -3.62 (25.96) | -4.55 (28.00)
  Role Functional Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 295
  Role Functional Scale: Change at Cycle 4 | -4.64 (27.69) | -5.99 (26.87)
  Role Functional Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Role Functional Scale: Change at Cycle 5 | -4.72 (27.68) | -7.41 (27.25)
  Role Functional Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Role Functional Scale: Change at Cycle 6 | -6.13 (28.94) | -6.03 (28.51)
  Role Functional Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 228
  Role Functional Scale: Change at Cycle 7 | -4.82 (29.75) | -5.34 (26.31)
  Role Functional Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Role Functional Scale: Change at Cycle 8 | -1.85 (28.87) | -2.38 (26.41)
  Role Functional Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Role Functional Scale: Change at Cycle 9 | -1.19 (28.57) | -2.47 (27.29)
  Role Functional Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Role Functional Scale: Change at Cycle 10 | -1.79 (28.10) | 0.90 (25.97)
  Role Functional Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Role Functional Scale: Change at Cycle 11 | -0.78 (28.34) | -2.69 (24.94)
  Role Functional Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Role Functional Scale: Change at Cycle 12 | -1.05 (27.28) | 0.24 (24.07)
  Role Functional Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Role Functional Scale: Change at Cycle 13 | -2.01 (26.61) | -2.40 (24.91)
  Role Functional Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Role Functional Scale: Change at Cycle 14 | -0.86 (27.27) | -1.31 (25.66)
  Role Functional Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Role Functional Scale: Change at Cycle 15 | -1.03 (27.51) | -3.23 (25.40)
  Role Functional Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Role Functional Scale: Change at Cycle 16 | -3.16 (28.73) | -2.35 (25.48)
  Role Functional Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Role Functional Scale: Change at Cycle 17 | -1.04 (26.69) | -3.38 (25.88)
  Role Functional Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Role Functional Scale: Change at Cycle 18 | -0.16 (27.10) | 0.23 (26.05)
  Role Functional Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Role Functional Scale: Change at Cycle 19 | 1.04 (27.55) | -0.25 (23.48)
  Role Functional Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Role Functional Scale: Change at Cycle 20 | -1.19 (30.04) | 0.79 (23.46)
  Role Functional Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Role Functional Scale: Change at Cycle 21 | -0.84 (28.98) | 0.00 (27.47)
  Role Functional Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Role Functional Scale: Change at Cycle 22 | -2.24 (27.96) | 1.06 (22.63)
  Role Functional Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Role Functional Scale: Change at Cycle 23 | -3.44 (30.11) | 1.14 (25.01)
  Role Functional Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Role Functional Scale: Change at Cycle 24 | -4.44 (29.73) | 2.08 (24.22)
  Role Functional Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Role Functional Scale: Change at Cycle 25 | -3.53 (29.21) | 4.63 (26.91)
  Role Functional Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Role Functional Scale: Change at Cycle 26 | -1.36 (28.02) | 0.52 (26.60)
  Role Functional Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Role Functional Scale: Change at Cycle 27 | -1.55 (30.82) | -4.02 (29.77)
  Role Functional Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Role Functional Scale: Change at Cycle 28 | -0.42 (27.86) | -3.85 (29.56)
  Role Functional Scale: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Role Functional Scale: Change at PT Visit 1 | -14.61 (30.41) | -9.49 (28.64)
  Role Functional Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Role Functional Scale: Change at PT Visit 2 | -10.73 (31.94) | -15.45 (31.82)
  Social Functional Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 381
  Social Functional Scale: Cycle 1 (Baseline) | 77.96 (24.09) | 75.90 (24.69)
  Social Functional Scale: Change at Cycle 2: number analyzed (Participants) | 333 | 341
  Social Functional Scale: Change at Cycle 2 | -3.45 (24.07) | -0.44 (23.09)
  Social Functional Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 314
  Social Functional Scale: Change at Cycle 3 | -4.62 (25.25) | -2.07 (25.35)
  Social Functional Scale: Change at Cycle 4: number analyzed (Participants) | 302 | 294
  Social Functional Scale: Change at Cycle 4 | -2.59 (25.08) | -1.70 (26.58)
  Social Functional Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 286
  Social Functional Scale: Change at Cycle 5 | -5.54 (27.03) | -3.26 (27.24)
  Social Functional Scale: Change at Cycle 6: number analyzed (Participants) | 271 | 256
  Social Functional Scale: Change at Cycle 6 | -5.72 (27.87) | -1.04 (27.20)
  Social Functional Scale: Change at Cycle 7: number analyzed (Participants) | 242 | 227
  Social Functional Scale: Change at Cycle 7 | -2.69 (27.13) | -0.15 (26.00)
  Social Functional Scale: Change at Cycle 8: number analyzed (Participants) | 233 | 216
  Social Functional Scale: Change at Cycle 8 | -1.72 (26.93) | 1.08 (26.49)
  Social Functional Scale: Change at Cycle 9: number analyzed (Participants) | 210 | 196
  Social Functional Scale: Change at Cycle 9 | 0.56 (27.59) | 0.77 (25.11)
  Social Functional Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Social Functional Scale: Change at Cycle 10 | -0.81 (27.31) | 2.31 (25.75)
  Social Functional Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Social Functional Scale: Change at Cycle 11 | 0.58 (27.35) | 1.94 (24.39)
  Social Functional Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 139
  Social Functional Scale: Change at Cycle 12 | 0.52 (28.59) | 2.40 (24.70)
  Social Functional Scale: Change at Cycle 13: number analyzed (Participants) | 140 | 111
  Social Functional Scale: Change at Cycle 13 | 0.83 (25.31) | 2.10 (25.73)
  Social Functional Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Social Functional Scale: Change at Cycle 14 | 1.98 (26.71) | 2.12 (24.89)
  Social Functional Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Social Functional Scale: Change at Cycle 15 | 1.79 (27.24) | 0.00 (27.08)
  Social Functional Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Social Functional Scale: Change at Cycle 16 | -0.72 (25.76) | 0.39 (25.84)
  Social Functional Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Social Functional Scale: Change at Cycle 17 | -0.45 (26.51) | 1.58 (24.39)
  Social Functional Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Social Functional Scale: Change at Cycle 18 | -0.98 (25.99) | 2.11 (26.42)
  Social Functional Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Social Functional Scale: Change at Cycle 19 | 2.26 (26.56) | 3.28 (21.53)
  Social Functional Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Social Functional Scale: Change at Cycle 20 | 1.59 (27.09) | 0.79 (22.88)
  Social Functional Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Social Functional Scale: Change at Cycle 21 | 1.27 (28.09) | 5.86 (22.00)
  Social Functional Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Social Functional Scale: Change at Cycle 22 | 1.24 (27.72) | 2.84 (24.16)
  Social Functional Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Social Functional Scale: Change at Cycle 23 | 6.08 (27.32) | 1.89 (22.51)
  Social Functional Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Social Functional Scale: Change at Cycle 24 | 5.83 (25.64) | 4.17 (24.39)
  Social Functional Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Social Functional Scale: Change at Cycle 25 | 1.60 (27.27) | 2.78 (23.40)
  Social Functional Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Social Functional Scale: Change at Cycle 26 | 3.74 (26.19) | 1.56 (24.45)
  Social Functional Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Social Functional Scale: Change at Cycle 27 | 5.81 (24.37) | -1.72 (26.85)
  Social Functional Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Social Functional Scale: Change at Cycle 28 | 6.25 (23.48) | -0.64 (24.26)
  Social Functional Scale: Change at PT Visit 1: number analyzed (Participants) | 177 | 202
  Social Functional Scale: Change at PT Visit 1 | -9.13 (26.47) | -3.80 (28.74)
  Social Functional Scale: Change at PT Visit 2: number analyzed (Participants) | 101 | 110
  Social Functional Scale: Change at PT Visit 2 | -5.45 (28.49) | -8.48 (28.98)
  Insomnia Symptom Scale: Cycle 1 (Baseline): number analyzed (Participants) | 372 | 383
  Insomnia Symptom Scale: Cycle 1 (Baseline) | 22.94 (28.00) | 25.41 (28.81)
  Insomnia Symptom Scale: Change at Cycle 2: number analyzed (Participants) | 336 | 343
  Insomnia Symptom Scale: Change at Cycle 2 | -0.69 (26.82) | -0.39 (28.27)
  Insomnia Symptom Scale: Change at Cycle 3: number analyzed (Participants) | 321 | 316
  Insomnia Symptom Scale: Change at Cycle 3 | -3.53 (27.03) | -3.48 (30.14)
  Insomnia Symptom Scale: Change at Cycle 4: number analyzed (Participants) | 301 | 295
  Insomnia Symptom Scale: Change at Cycle 4 | -2.88 (28.14) | -3.62 (30.40)
  Insomnia Symptom Scale: Change at Cycle 5: number analyzed (Participants) | 286 | 288
  Insomnia Symptom Scale: Change at Cycle 5 | -2.21 (29.27) | -2.66 (30.17)
  Insomnia Symptom Scale: Change at Cycle 6: number analyzed (Participants) | 272 | 257
  Insomnia Symptom Scale: Change at Cycle 6 | -2.94 (28.63) | -5.58 (32.53)
  Insomnia Symptom Scale: Change at Cycle 7: number analyzed (Participants) | 241 | 228
  Insomnia Symptom Scale: Change at Cycle 7 | -4.56 (28.42) | -4.82 (32.98)
  Insomnia Symptom Scale: Change at Cycle 8: number analyzed (Participants) | 234 | 217
  Insomnia Symptom Scale: Change at Cycle 8 | -6.13 (27.72) | -6.45 (30.75)
  Insomnia Symptom Scale: Change at Cycle 9: number analyzed (Participants) | 208 | 196
  Insomnia Symptom Scale: Change at Cycle 9 | -8.97 (25.69) | -6.12 (30.32)
  Insomnia Symptom Scale: Change at Cycle 10: number analyzed (Participants) | 186 | 166
  Insomnia Symptom Scale: Change at Cycle 10 | -8.24 (26.69) | -4.42 (28.79)
  Insomnia Symptom Scale: Change at Cycle 11: number analyzed (Participants) | 171 | 155
  Insomnia Symptom Scale: Change at Cycle 11 | -8.97 (28.19) | -5.81 (27.69)
  Insomnia Symptom Scale: Change at Cycle 12: number analyzed (Participants) | 159 | 140
  Insomnia Symptom Scale: Change at Cycle 12 | -8.81 (27.67) | -6.43 (26.49)
  Insomnia Symptom Scale: Change at Cycle 13: number analyzed (Participants) | 141 | 111
  Insomnia Symptom Scale: Change at Cycle 13 | -10.17 (26.71) | -5.11 (24.29)
  Insomnia Symptom Scale: Change at Cycle 14: number analyzed (Participants) | 135 | 102
  Insomnia Symptom Scale: Change at Cycle 14 | -9.14 (26.84) | -7.84 (24.45)
  Insomnia Symptom Scale: Change at Cycle 15: number analyzed (Participants) | 130 | 98
  Insomnia Symptom Scale: Change at Cycle 15 | -9.74 (28.89) | -5.10 (21.59)
  Insomnia Symptom Scale: Change at Cycle 16: number analyzed (Participants) | 116 | 85
  Insomnia Symptom Scale: Change at Cycle 16 | -8.91 (26.14) | -4.31 (26.62)
  Insomnia Symptom Scale: Change at Cycle 17: number analyzed (Participants) | 112 | 74
  Insomnia Symptom Scale: Change at Cycle 17 | -11.01 (26.62) | -5.41 (26.48)
  Insomnia Symptom Scale: Change at Cycle 18: number analyzed (Participants) | 102 | 71
  Insomnia Symptom Scale: Change at Cycle 18 | -8.82 (28.12) | -8.45 (20.09)
  Insomnia Symptom Scale: Change at Cycle 19: number analyzed (Participants) | 96 | 66
  Insomnia Symptom Scale: Change at Cycle 19 | -11.46 (29.35) | -7.58 (22.49)
  Insomnia Symptom Scale: Change at Cycle 20: number analyzed (Participants) | 84 | 63
  Insomnia Symptom Scale: Change at Cycle 20 | -10.32 (27.37) | -5.29 (25.55)
  Insomnia Symptom Scale: Change at Cycle 21: number analyzed (Participants) | 79 | 54
  Insomnia Symptom Scale: Change at Cycle 21 | -11.81 (27.24) | -4.94 (27.02)
  Insomnia Symptom Scale: Change at Cycle 22: number analyzed (Participants) | 67 | 47
  Insomnia Symptom Scale: Change at Cycle 22 | -10.95 (31.46) | -7.80 (19.92)
  Insomnia Symptom Scale: Change at Cycle 23: number analyzed (Participants) | 63 | 44
  Insomnia Symptom Scale: Change at Cycle 23 | -10.58 (34.82) | -6.06 (23.04)
  Insomnia Symptom Scale: Change at Cycle 24: number analyzed (Participants) | 60 | 40
  Insomnia Symptom Scale: Change at Cycle 24 | -9.44 (31.94) | -7.50 (21.99)
  Insomnia Symptom Scale: Change at Cycle 25: number analyzed (Participants) | 52 | 36
  Insomnia Symptom Scale: Change at Cycle 25 | -10.26 (28.42) | -8.33 (26.87)
  Insomnia Symptom Scale: Change at Cycle 26: number analyzed (Participants) | 49 | 32
  Insomnia Symptom Scale: Change at Cycle 26 | -9.52 (32.63) | -4.17 (20.30)
  Insomnia Symptom Scale: Change at Cycle 27: number analyzed (Participants) | 43 | 29
  Insomnia Symptom Scale: Change at Cycle 27 | -13.18 (30.11) | -4.60 (19.36)
  Insomnia Symptom Scale: Change at Cycle 28: number analyzed (Participants) | 40 | 26
  Insomnia Symptom Scale: Change at Cycle 28 | -11.67 (31.62) | -1.28 (22.07)
  Insomnia Symptom Scale: Change at PT Visit 1: number analyzed (Participants) | 178 | 202
  Insomnia Symptom Scale: Change at PT Visit 1 | 2.81 (29.19) | -1.32 (30.81)
  Insomnia Symptom Scale: Change at PT Visit 2: number analyzed (Participants) | 100 | 110
  Insomnia Symptom Scale: Change at PT Visit 2 | 5.67 (29.23) | 3.03 (31.13)

10. Secondary Outcome: Change From Baseline in EORTC QLQ-Gastric Cancer Module (EORTC QLQ-STO22) Score
Description: The EORTC QLQ-STO22 is a gastric cancer quality of life questionnaire. There are 22 questions concerning disease, treatment related symptoms, side effects, dysphagia, nutritional aspects, and questions about the emotional problems of gastric cancer (dysphagia, pain, reflux, eating restrictions, anxiety, dry mouth, body image, and hair loss). The questions are grouped into five scales and 4 single items which are related to the symptoms of the disease. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms. A positive value means an increase, while a negative values means a decrease, in score at the indicated time-point relative to the score at baseline (Cycle 1, Day 1).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 388 | 392
score on a scale
  Anxiety: Cycle 1 (Baseline): number analyzed (Participants) | 366 | 373
  Anxiety: Cycle 1 (Baseline) | 40.10 (25.85) | 40.48 (25.32)
  Anxiety: Change at Cycle 2: number analyzed (Participants) | 329 | 334
  Anxiety: Change at Cycle 2 | -2.58 (21.72) | -4.11 (21.19)
  Anxiety: Change at Cycle 3: number analyzed (Participants) | 317 | 309
  Anxiety: Change at Cycle 3 | -4.14 (22.45) | -3.87 (23.19)
  Anxiety: Change at Cycle 4: number analyzed (Participants) | 295 | 289
  Anxiety: Change at Cycle 4 | -4.52 (23.01) | -7.25 (23.16)
  Anxiety: Change at Cycle 5: number analyzed (Participants) | 282 | 285
  Anxiety: Change at Cycle 5 | -4.10 (22.94) | -7.39 (24.36)
  Anxiety: Change at Cycle 6: number analyzed (Participants) | 269 | 252
  Anxiety: Change at Cycle 6 | -4.54 (23.97) | -8.42 (25.21)
  Anxiety: Change at Cycle 7: number analyzed (Participants) | 238 | 226
  Anxiety: Change at Cycle 7 | -6.40 (24.00) | -10.40 (24.37)
  Anxiety: Change at Cycle 8: number analyzed (Participants) | 232 | 213
  Anxiety: Change at Cycle 8 | -9.00 (23.17) | -11.92 (24.50)
  Anxiety: Change at Cycle 9: number analyzed (Participants) | 206 | 193
  Anxiety: Change at Cycle 9 | -10.09 (23.30) | -11.43 (23.24)
  Anxiety: Change at Cycle 10: number analyzed (Participants) | 185 | 164
  Anxiety: Change at Cycle 10 | -11.17 (25.05) | -12.64 (22.09)
  Anxiety: Change at Cycle 11: number analyzed (Participants) | 168 | 153
  Anxiety: Change at Cycle 11 | -10.78 (23.47) | -12.09 (21.84)
  Anxiety: Change at Cycle 12: number analyzed (Participants) | 158 | 138
  Anxiety: Change at Cycle 12 | -12.62 (26.24) | -13.16 (23.11)
  Anxiety: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Anxiety: Change at Cycle 13 | -13.32 (25.93) | -13.33 (22.47)
  Anxiety: Change at Cycle 14: number analyzed (Participants) | 135 | 101
  Anxiety: Change at Cycle 14 | -14.32 (26.49) | -12.43 (23.59)
  Anxiety: Change at Cycle 15: number analyzed (Participants) | 130 | 96
  Anxiety: Change at Cycle 15 | -13.42 (26.64) | -10.65 (25.74)
  Anxiety: Change at Cycle 16: number analyzed (Participants) | 115 | 84
  Anxiety: Change at Cycle 16 | -12.75 (26.87) | -12.57 (23.89)
  Anxiety: Change at Cycle 17: number analyzed (Participants) | 111 | 73
  Anxiety: Change at Cycle 17 | -13.41 (27.30) | -12.79 (21.01)
  Anxiety: Change at Cycle 18: number analyzed (Participants) | 101 | 70
  Anxiety: Change at Cycle 18 | -13.53 (28.05) | -12.38 (22.90)
  Anxiety: Change at Cycle 19: number analyzed (Participants) | 95 | 65
  Anxiety: Change at Cycle 19 | -14.50 (27.41) | -12.48 (20.08)
  Anxiety: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Anxiety: Change at Cycle 20 | -15.34 (29.21) | -12.37 (23.73)
  Anxiety: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Anxiety: Change at Cycle 21 | -16.03 (28.84) | -14.47 (25.00)
  Anxiety: Change at Cycle 22: number analyzed (Participants) | 66 | 46
  Anxiety: Change at Cycle 22 | -13.30 (30.77) | -15.46 (23.83)
  Anxiety: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Anxiety: Change at Cycle 23 | -17.28 (30.64) | -14.47 (29.55)
  Anxiety: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Anxiety: Change at Cycle 24 | -16.11 (30.65) | -17.09 (23.76)
  Anxiety: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Anxiety: Change at Cycle 25 | -16.03 (29.47) | -17.78 (23.68)
  Anxiety: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Anxiety: Change at Cycle 26 | -19.73 (30.28) | -13.26 (22.11)
  Anxiety: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Anxiety: Change at Cycle 27 | -21.71 (29.89) | -12.70 (20.67)
  Anxiety: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Anxiety: Change at Cycle 28 | -22.51 (29.34) | -12.89 (22.38)
  Anxiety: Change at PT Visit 1: number analyzed (Participants) | 175 | 196
  Anxiety: Change at PT Visit 1 | -0.73 (25.18) | -4.73 (27.21)
  Anxiety: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Anxiety: Change at PT Visit 2 | -4.04 (28.24) | -3.98 (25.02)
  Body Image: Cycle 1 (Baseline): number analyzed (Participants) | 364 | 373
  Body Image: Cycle 1 (Baseline) | 23.53 (28.40) | 23.68 (27.47)
  Body Image: Change at Cycle 2: number analyzed (Participants) | 326 | 334
  Body Image: Change at Cycle 2 | 1.33 (28.19) | 1.20 (26.44)
  Body Image: Change at Cycle 3: number analyzed (Participants) | 316 | 309
  Body Image: Change at Cycle 3 | 1.48 (29.06) | 3.88 (28.03)
  Body Image: Change at Cycle 4: number analyzed (Participants) | 294 | 289
  Body Image: Change at Cycle 4 | 4.20 (28.51) | 1.15 (27.19)
  Body Image: Change at Cycle 5: number analyzed (Participants) | 280 | 284
  Body Image: Change at Cycle 5 | 2.86 (30.91) | 1.06 (25.74)
  Body Image: Change at Cycle 6: number analyzed (Participants) | 268 | 252
  Body Image: Change at Cycle 6 | 0.75 (30.11) | 2.78 (28.48)
  Body Image: Change at Cycle 7: number analyzed (Participants) | 237 | 226
  Body Image: Change at Cycle 7 | -0.56 (28.94) | 0.29 (25.53)
  Body Image: Change at Cycle 8: number analyzed (Participants) | 230 | 213
  Body Image: Change at Cycle 8 | -1.74 (29.83) | 0.00 (26.30)
  Body Image: Change at Cycle 9: number analyzed (Participants) | 205 | 193
  Body Image: Change at Cycle 9 | -3.58 (28.74) | -0.69 (24.52)
  Body Image: Change at Cycle 10: number analyzed (Participants) | 184 | 164
  Body Image: Change at Cycle 10 | -5.07 (30.15) | -3.25 (24.55)
  Body Image: Change at Cycle 11: number analyzed (Participants) | 166 | 153
  Body Image: Change at Cycle 11 | -4.62 (30.24) | -1.53 (25.46)
  Body Image: Change at Cycle 12: number analyzed (Participants) | 157 | 138
  Body Image: Change at Cycle 12 | -5.31 (31.92) | -2.66 (27.04)
  Body Image: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Body Image: Change at Cycle 13 | -4.73 (30.23) | -2.73 (25.99)
  Body Image: Change at Cycle 14: number analyzed (Participants) | 135 | 101
  Body Image: Change at Cycle 14 | -5.43 (29.70) | -4.62 (24.05)
  Body Image: Change at Cycle 15: number analyzed (Participants) | 130 | 96
  Body Image: Change at Cycle 15 | -3.08 (30.63) | -2.43 (27.03)
  Body Image: Change at Cycle 16: number analyzed (Participants) | 115 | 84
  Body Image: Change at Cycle 16 | -1.74 (32.99) | -1.19 (26.10)
  Body Image: Change at Cycle 17: number analyzed (Participants) | 111 | 73
  Body Image: Change at Cycle 17 | -2.70 (32.76) | -2.28 (21.75)
  Body Image: Change at Cycle 18: number analyzed (Participants) | 101 | 70
  Body Image: Change at Cycle 18 | -2.64 (30.44) | -5.71 (23.38)
  Body Image: Change at Cycle 19: number analyzed (Participants) | 95 | 64
  Body Image: Change at Cycle 19 | -2.81 (33.57) | -5.21 (20.76)
  Body Image: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Body Image: Change at Cycle 20 | -3.97 (30.79) | -5.38 (22.74)
  Body Image: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Body Image: Change at Cycle 21 | 1.69 (30.15) | -8.18 (26.07)
  Body Image: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Body Image: Change at Cycle 22 | -1.49 (32.01) | -10.87 (22.28)
  Body Image: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Body Image: Change at Cycle 23 | -5.82 (24.35) | -8.53 (29.18)
  Body Image: Change at Cycle 24: number analyzed (Participants) | 59 | 39
  Body Image: Change at Cycle 24 | -0.56 (31.25) | -11.11 (23.36)
  Body Image: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Body Image: Change at Cycle 25 | -3.21 (28.97) | -11.43 (24.18)
  Body Image: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Body Image: Change at Cycle 26 | -4.76 (29.66) | -6.45 (18.09)
  Body Image: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Body Image: Change at Cycle 27 | 0.78 (24.65) | -7.14 (21.00)
  Body Image: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Body Image: Change at Cycle 28 | -4.27 (26.69) | -4.00 (24.19)
  Body Image: Change at PT Visit 1: number analyzed (Participants) | 175 | 195
  Body Image: Change at PT Visit 1 | 2.48 (31.57) | 3.42 (29.31)
  Body Image: Change at PT Visit 2: number analyzed (Participants) | 99 | 105
  Body Image: Change at PT Visit 2 | 2.36 (35.40) | 6.35 (27.38)
  Dry Mouth: Cycle 1 (Baseline): number analyzed (Participants) | 367 | 373
  Dry Mouth: Cycle 1 (Baseline) | 21.80 (25.07) | 23.32 (26.79)
  Dry Mouth: Change at Cycle 2: number analyzed (Participants) | 328 | 333
  Dry Mouth: Change at Cycle 2 | 7.72 (28.70) | 3.00 (25.43)
  Dry Mouth: Change at Cycle 3: number analyzed (Participants) | 317 | 308
  Dry Mouth: Change at Cycle 3 | 6.10 (28.65) | 4.87 (27.33)
  Dry Mouth: Change at Cycle 4: number analyzed (Participants) | 294 | 288
  Dry Mouth: Change at Cycle 4 | 4.76 (29.40) | 2.66 (31.06)
  Dry Mouth: Change at Cycle 5: number analyzed (Participants) | 283 | 285
  Dry Mouth: Change at Cycle 5 | 2.47 (29.67) | 2.57 (28.68)
  Dry Mouth: Change at Cycle 6: number analyzed (Participants) | 270 | 252
  Dry Mouth: Change at Cycle 6 | 2.96 (30.14) | 1.19 (27.65)
  Dry Mouth: Change at Cycle 7: number analyzed (Participants) | 238 | 226
  Dry Mouth: Change at Cycle 7 | -1.96 (28.82) | 0.44 (28.54)
  Dry Mouth: Change at Cycle 8: number analyzed (Participants) | 233 | 213
  Dry Mouth: Change at Cycle 8 | -2.43 (28.68) | -2.66 (26.27)
  Dry Mouth: Change at Cycle 9: number analyzed (Participants) | 207 | 193
  Dry Mouth: Change at Cycle 9 | -3.70 (25.70) | -4.32 (24.74)
  Dry Mouth: Change at Cycle 10: number analyzed (Participants) | 186 | 164
  Dry Mouth: Change at Cycle 10 | -6.27 (25.04) | -3.46 (23.53)
  Dry Mouth: Change at Cycle 11: number analyzed (Participants) | 169 | 153
  Dry Mouth: Change at Cycle 11 | -7.69 (25.46) | -1.96 (26.56)
  Dry Mouth: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Dry Mouth: Change at Cycle 12 | -8.18 (24.22) | -4.35 (26.36)
  Dry Mouth: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Dry Mouth: Change at Cycle 13 | -9.69 (24.08) | -8.48 (26.50)
  Dry Mouth: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Dry Mouth: Change at Cycle 14 | -8.33 (24.60) | -3.63 (29.78)
  Dry Mouth: Change at Cycle 15: number analyzed (Participants) | 131 | 96
  Dry Mouth: Change at Cycle 15 | -7.89 (22.20) | -7.29 (26.58)
  Dry Mouth: Change at Cycle 16: number analyzed (Participants) | 116 | 84
  Dry Mouth: Change at Cycle 16 | -6.32 (24.44) | -8.33 (27.80)
  Dry Mouth: Change at Cycle 17: number analyzed (Participants) | 112 | 73
  Dry Mouth: Change at Cycle 17 | -7.44 (23.12) | -3.20 (24.32)
  Dry Mouth: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Dry Mouth: Change at Cycle 18 | -5.56 (24.86) | -8.10 (28.62)
  Dry Mouth: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Dry Mouth: Change at Cycle 19 | -5.90 (24.18) | -7.69 (25.53)
  Dry Mouth: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Dry Mouth: Change at Cycle 20 | -6.35 (26.62) | -9.68 (27.25)
  Dry Mouth: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Dry Mouth: Change at Cycle 21 | -7.17 (24.27) | -9.43 (20.02)
  Dry Mouth: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Dry Mouth: Change at Cycle 22 | -3.98 (26.29) | -8.70 (23.76)
  Dry Mouth: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Dry Mouth: Change at Cycle 23 | -7.94 (23.73) | -3.88 (25.42)
  Dry Mouth: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Dry Mouth: Change at Cycle 24 | -6.67 (25.15) | -9.40 (28.56)
  Dry Mouth: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Dry Mouth: Change at Cycle 25 | -8.33 (22.75) | -9.52 (28.66)
  Dry Mouth: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Dry Mouth: Change at Cycle 26 | -2.72 (23.41) | -7.53 (26.82)
  Dry Mouth: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Dry Mouth: Change at Cycle 27 | -6.98 (21.28) | -7.14 (27.75)
  Dry Mouth: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Dry Mouth: Change at Cycle 28 | -8.55 (21.24) | -8.00 (22.11)
  Dry Mouth: Change at PT Visit 1: number analyzed (Participants) | 175 | 196
  Dry Mouth: Change at PT Visit 1 | 0.19 (28.70) | 2.38 (31.58)
  Dry Mouth: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Dry Mouth: Change at PT Visit 2 | -1.35 (30.09) | 1.89 (25.95)
  Dysphagia: Cycle 1 (Baseline): number analyzed (Participants) | 367 | 373
  Dysphagia: Cycle 1 (Baseline) | 16.29 (21.46) | 14.15 (18.93)
  Dysphagia: Change at Cycle 2: number analyzed (Participants) | 330 | 334
  Dysphagia: Change at Cycle 2 | -2.27 (17.64) | -0.53 (19.32)
  Dysphagia: Change at Cycle 3: number analyzed (Participants) | 318 | 308
  Dysphagia: Change at Cycle 3 | -3.39 (18.57) | -2.15 (19.67)
  Dysphagia: Change at Cycle 4: number analyzed (Participants) | 295 | 289
  Dysphagia: Change at Cycle 4 | -2.94 (18.93) | -1.08 (18.79)
  Dysphagia: Change at Cycle 5: number analyzed (Participants) | 283 | 285
  Dysphagia: Change at Cycle 5 | -3.22 (19.92) | -1.83 (18.99)
  Dysphagia: Change at Cycle 6: number analyzed (Participants) | 270 | 252
  Dysphagia: Change at Cycle 6 | -4.20 (18.99) | -2.25 (18.70)
  Dysphagia: Change at Cycle 7: number analyzed (Participants) | 239 | 226
  Dysphagia: Change at Cycle 7 | -4.83 (20.56) | -1.97 (19.94)
  Dysphagia: Change at Cycle 8: number analyzed (Participants) | 233 | 213
  Dysphagia: Change at Cycle 8 | -5.96 (18.80) | -3.29 (18.48)
  Dysphagia: Change at Cycle 9: number analyzed (Participants) | 207 | 193
  Dysphagia: Change at Cycle 9 | -6.17 (18.21) | -3.86 (18.49)
  Dysphagia: Change at Cycle 10: number analyzed (Participants) | 186 | 164
  Dysphagia: Change at Cycle 10 | -6.03 (17.37) | -4.61 (16.87)
  Dysphagia: Change at Cycle 11: number analyzed (Participants) | 169 | 153
  Dysphagia: Change at Cycle 11 | -6.25 (17.09) | -2.83 (17.03)
  Dysphagia: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Dysphagia: Change at Cycle 12 | -7.06 (17.65) | -4.19 (15.84)
  Dysphagia: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Dysphagia: Change at Cycle 13 | -6.93 (18.71) | -3.54 (17.61)
  Dysphagia: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Dysphagia: Change at Cycle 14 | -8.01 (18.53) | -4.95 (18.22)
  Dysphagia: Change at Cycle 15: number analyzed (Participants) | 131 | 96
  Dysphagia: Change at Cycle 15 | -6.45 (17.38) | -2.14 (18.69)
  Dysphagia: Change at Cycle 16: number analyzed (Participants) | 116 | 84
  Dysphagia: Change at Cycle 16 | -4.41 (18.29) | -3.70 (21.08)
  Dysphagia: Change at Cycle 17: number analyzed (Participants) | 112 | 73
  Dysphagia: Change at Cycle 17 | -5.36 (16.87) | -3.20 (14.99)
  Dysphagia: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Dysphagia: Change at Cycle 18 | -4.90 (16.44) | -3.33 (19.78)
  Dysphagia: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Dysphagia: Change at Cycle 19 | -4.40 (17.10) | -3.59 (14.31)
  Dysphagia: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Dysphagia: Change at Cycle 20 | -2.51 (16.21) | -3.76 (15.83)
  Dysphagia: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Dysphagia: Change at Cycle 21 | -3.80 (19.24) | -2.10 (17.84)
  Dysphagia: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Dysphagia: Change at Cycle 22 | -3.65 (20.41) | -4.83 (15.65)
  Dysphagia: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Dysphagia: Change at Cycle 23 | -4.23 (18.87) | -3.88 (17.63)
  Dysphagia: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Dysphagia: Change at Cycle 24 | -5.00 (18.35) | -3.70 (13.08)
  Dysphagia: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Dysphagia: Change at Cycle 25 | -5.98 (19.61) | -2.22 (16.79)
  Dysphagia: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Dysphagia: Change at Cycle 26 | -5.67 (20.43) | -2.87 (16.22)
  Dysphagia: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Dysphagia: Change at Cycle 27 | -5.68 (20.91) | -4.37 (12.22)
  Dysphagia: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Dysphagia: Change at Cycle 28 | -8.26 (19.86) | -3.56 (11.44)
  Dysphagia: Change at PT Visit 1: number analyzed (Participants) | 176 | 196
  Dysphagia: Change at PT Visit 1 | 0.44 (24.15) | 2.83 (22.63)
  Dysphagia: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Dysphagia: Change at PT Visit 2 | -2.81 (24.40) | 3.25 (19.81)
  Eating Restrictions: Cycle 1 (Baseline): number analyzed (Participants) | 366 | 373
  Eating Restrictions: Cycle 1 (Baseline) | 23.26 (21.78) | 22.33 (20.22)
  Eating Restrictions: Change at Cycle 2: number analyzed (Participants) | 328 | 334
  Eating Restrictions: Change at Cycle 2 | -1.41 (19.36) | -1.54 (19.62)
  Eating Restrictions: Change at Cycle 3: number analyzed (Participants) | 318 | 308
  Eating Restrictions: Change at Cycle 3 | -1.04 (21.09) | -2.20 (20.94)
  Eating Restrictions: Change at Cycle 4: number analyzed (Participants) | 295 | 289
  Eating Restrictions: Change at Cycle 4 | -2.24 (20.81) | -1.39 (23.36)
  Eating Restrictions: Change at Cycle 5: number analyzed (Participants) | 283 | 285
  Eating Restrictions: Change at Cycle 5 | -1.39 (22.10) | -0.09 (23.31)
  Eating Restrictions: Change at Cycle 6: number analyzed (Participants) | 270 | 252
  Eating Restrictions: Change at Cycle 6 | -1.35 (22.77) | -3.32 (23.14)
  Eating Restrictions: Change at Cycle 7: number analyzed (Participants) | 239 | 225
  Eating Restrictions: Change at Cycle 7 | -2.45 (22.68) | -2.67 (21.66)
  Eating Restrictions: Change at Cycle 8: number analyzed (Participants) | 233 | 213
  Eating Restrictions: Change at Cycle 8 | -4.29 (22.70) | -5.56 (19.87)
  Eating Restrictions: Change at Cycle 9: number analyzed (Participants) | 207 | 193
  Eating Restrictions: Change at Cycle 9 | -6.99 (21.16) | -6.48 (19.69)
  Eating Restrictions: Change at Cycle 10: number analyzed (Participants) | 186 | 164
  Eating Restrictions: Change at Cycle 10 | -7.06 (21.32) | -5.89 (19.30)
  Eating Restrictions: Change at Cycle 11: number analyzed (Participants) | 169 | 153
  Eating Restrictions: Change at Cycle 11 | -8.22 (21.25) | -5.05 (19.98)
  Eating Restrictions: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Eating Restrictions: Change at Cycle 12 | -7.74 (21.16) | -6.34 (19.87)
  Eating Restrictions: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Eating Restrictions: Change at Cycle 13 | -8.55 (20.41) | -8.41 (19.57)
  Eating Restrictions: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Eating Restrictions: Change at Cycle 14 | -8.62 (19.16) | -8.58 (21.16)
  Eating Restrictions: Change at Cycle 15: number analyzed (Participants) | 131 | 96
  Eating Restrictions: Change at Cycle 15 | -6.85 (20.92) | -5.56 (21.21)
  Eating Restrictions: Change at Cycle 16: number analyzed (Participants) | 116 | 84
  Eating Restrictions: Change at Cycle 16 | -5.77 (22.01) | -6.94 (20.36)
  Eating Restrictions: Change at Cycle 17: number analyzed (Participants) | 112 | 73
  Eating Restrictions: Change at Cycle 17 | -5.56 (21.95) | -7.42 (17.76)
  Eating Restrictions: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Eating Restrictions: Change at Cycle 18 | -7.27 (20.40) | -6.90 (21.14)
  Eating Restrictions: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Eating Restrictions: Change at Cycle 19 | -7.03 (21.78) | -5.38 (18.07)
  Eating Restrictions: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Eating Restrictions: Change at Cycle 20 | -4.56 (21.03) | -4.44 (16.72)
  Eating Restrictions: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Eating Restrictions: Change at Cycle 21 | -5.80 (22.58) | -5.03 (19.97)
  Eating Restrictions: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Eating Restrictions: Change at Cycle 22 | -3.65 (21.79) | -6.16 (16.80)
  Eating Restrictions: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Eating Restrictions: Change at Cycle 23 | -3.70 (22.74) | -5.23 (20.25)
  Eating Restrictions: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Eating Restrictions: Change at Cycle 24 | -5.00 (20.77) | -7.91 (15.76)
  Eating Restrictions: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Eating Restrictions: Change at Cycle 25 | -5.77 (21.10) | -5.95 (16.61)
  Eating Restrictions: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Eating Restrictions: Change at Cycle 26 | -6.80 (21.22) | -2.42 (22.89)
  Eating Restrictions: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Eating Restrictions: Change at Cycle 27 | -5.62 (23.48) | -3.87 (10.26)
  Eating Restrictions: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Eating Restrictions: Change at Cycle 28 | -7.91 (21.79) | -5.00 (11.02)
  Eating Restrictions: Change at PT Visit 1: number analyzed (Participants) | 176 | 196
  Eating Restrictions: Change at PT Visit 1 | 1.52 (24.48) | 0.94 (24.70)
  Eating Restrictions: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Eating Restrictions: Change at PT Visit 2 | -2.10 (25.32) | 0.94 (21.46)
  Hair Loss: Cycle 1 (Baseline): number analyzed (Participants) | 363 | 371
  Hair Loss: Cycle 1 (Baseline) | 4.73 (13.28) | 4.04 (13.20)
  Hair Loss: Change at Cycle 2: number analyzed (Participants) | 326 | 329
  Hair Loss: Change at Cycle 2 | 0.20 (14.85) | 1.27 (16.59)
  Hair Loss: Change at Cycle 3: number analyzed (Participants) | 315 | 306
  Hair Loss: Change at Cycle 3 | 4.34 (17.51) | 4.52 (18.71)
  Hair Loss: Change at Cycle 4: number analyzed (Participants) | 293 | 286
  Hair Loss: Change at Cycle 4 | 5.40 (18.46) | 6.53 (20.99)
  Hair Loss: Change at Cycle 5: number analyzed (Participants) | 278 | 281
  Hair Loss: Change at Cycle 5 | 6.12 (19.38) | 7.18 (19.49)
  Hair Loss: Change at Cycle 6: number analyzed (Participants) | 267 | 250
  Hair Loss: Change at Cycle 6 | 6.93 (18.87) | 10.07 (22.94)
  Hair Loss: Change at Cycle 7: number analyzed (Participants) | 236 | 225
  Hair Loss: Change at Cycle 7 | 5.72 (19.91) | 9.26 (22.92)
  Hair Loss: Change at Cycle 8: number analyzed (Participants) | 230 | 210
  Hair Loss: Change at Cycle 8 | 5.00 (18.96) | 7.38 (23.05)
  Hair Loss: Change at Cycle 9: number analyzed (Participants) | 203 | 191
  Hair Loss: Change at Cycle 9 | 2.38 (17.43) | 6.46 (21.06)
  Hair Loss: Change at Cycle 10: number analyzed (Participants) | 183 | 162
  Hair Loss: Change at Cycle 10 | 0.64 (16.88) | 4.22 (19.51)
  Hair Loss: Change at Cycle 11: number analyzed (Participants) | 165 | 151
  Hair Loss: Change at Cycle 11 | -0.10 (17.02) | 2.54 (17.51)
  Hair Loss: Change at Cycle 12: number analyzed (Participants) | 157 | 136
  Hair Loss: Change at Cycle 12 | 0.21 (19.70) | 1.96 (15.72)
  Hair Loss: Change at Cycle 13: number analyzed (Participants) | 140 | 109
  Hair Loss: Change at Cycle 13 | 0.36 (18.91) | 2.29 (15.46)
  Hair Loss: Change at Cycle 14: number analyzed (Participants) | 134 | 100
  Hair Loss: Change at Cycle 14 | -1.37 (17.59) | 1.83 (15.15)
  Hair Loss: Change at Cycle 15: number analyzed (Participants) | 129 | 95
  Hair Loss: Change at Cycle 15 | -0.39 (15.65) | 1.58 (12.65)
  Hair Loss: Change at Cycle 16: number analyzed (Participants) | 113 | 82
  Hair Loss: Change at Cycle 16 | -1.47 (17.47) | 1.42 (13.91)
  Hair Loss: Change at Cycle 17: number analyzed (Participants) | 109 | 73
  Hair Loss: Change at Cycle 17 | -1.07 (17.75) | 0.23 (12.57)
  Hair Loss: Change at Cycle 18: number analyzed (Participants) | 99 | 70
  Hair Loss: Change at Cycle 18 | -1.68 (17.58) | -0.71 (13.14)
  Hair Loss: Change at Cycle 19: number analyzed (Participants) | 93 | 65
  Hair Loss: Change at Cycle 19 | -0.90 (18.12) | 0.51 (14.12)
  Hair Loss: Change at Cycle 20: number analyzed (Participants) | 83 | 62
  Hair Loss: Change at Cycle 20 | -0.20 (19.21) | -1.61 (12.70)
  Hair Loss: Change at Cycle 21: number analyzed (Participants) | 78 | 53
  Hair Loss: Change at Cycle 21 | -1.07 (19.43) | -1.57 (8.81)
  Hair Loss: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Hair Loss: Change at Cycle 22 | -0.50 (16.66) | -3.26 (11.98)
  Hair Loss: Change at Cycle 23: number analyzed (Participants) | 62 | 42
  Hair Loss: Change at Cycle 23 | -0.54 (16.79) | -1.19 (11.28)
  Hair Loss: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Hair Loss: Change at Cycle 24 | -1.39 (17.44) | 1.71 (16.13)
  Hair Loss: Change at Cycle 25: number analyzed (Participants) | 51 | 35
  Hair Loss: Change at Cycle 25 | -1.96 (18.75) | -0.95 (9.85)
  Hair Loss: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Hair Loss: Change at Cycle 26 | -1.02 (19.37) | -0.54 (10.08)
  Hair Loss: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Hair Loss: Change at Cycle 27 | -3.10 (15.96) | -0.60 (10.62)
  Hair Loss: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Hair Loss: Change at Cycle 28 | -4.70 (20.57) | -1.33 (10.67)
  Hair Loss: Change at PT Visit 1: number analyzed (Participants) | 174 | 192
  Hair Loss: Change at PT Visit 1 | 4.98 (19.73) | 4.51 (20.39)
  Hair Loss: Change at PT Visit 2: number analyzed (Participants) | 99 | 105
  Hair Loss: Change at PT Visit 2 | 15.82 (25.35) | 22.22 (30.81)
  Pain: Cycle 1 (Baseline): number analyzed (Participants) | 367 | 373
  Pain: Cycle 1 (Baseline) | 26.48 (21.34) | 26.47 (20.70)
  Pain: Change at Cycle 2: number analyzed (Participants) | 330 | 334
  Pain: Change at Cycle 2 | -4.63 (20.30) | -5.86 (19.15)
  Pain: Change at Cycle 3: number analyzed (Participants) | 318 | 308
  Pain: Change at Cycle 3 | -6.96 (20.37) | -5.86 (20.68)
  Pain: Change at Cycle 4: number analyzed (Participants) | 296 | 289
  Pain: Change at Cycle 4 | -6.45 (21.47) | -7.48 (21.23)
  Pain: Change at Cycle 5: number analyzed (Participants) | 283 | 285
  Pain: Change at Cycle 5 | -7.28 (20.95) | -6.89 (22.10)
  Pain: Change at Cycle 6: number analyzed (Participants) | 270 | 252
  Pain: Change at Cycle 6 | -7.24 (20.84) | -7.22 (21.62)
  Pain: Change at Cycle 7: number analyzed (Participants) | 239 | 226
  Pain: Change at Cycle 7 | -9.52 (21.18) | -6.62 (21.63)
  Pain: Change at Cycle 8: number analyzed (Participants) | 233 | 213
  Pain: Change at Cycle 8 | -10.53 (21.62) | -8.16 (20.11)
  Pain: Change at Cycle 9: number analyzed (Participants) | 207 | 193
  Pain: Change at Cycle 9 | -10.08 (19.60) | -8.98 (20.29)
  Pain: Change at Cycle 10: number analyzed (Participants) | 186 | 164
  Pain: Change at Cycle 10 | -10.63 (19.23) | -8.59 (20.38)
  Pain: Change at Cycle 11: number analyzed (Participants) | 169 | 153
  Pain: Change at Cycle 11 | -11.65 (19.35) | -8.01 (18.97)
  Pain: Change at Cycle 12: number analyzed (Participants) | 159 | 138
  Pain: Change at Cycle 12 | -11.76 (19.87) | -7.19 (19.11)
  Pain: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Pain: Change at Cycle 13 | -11.92 (18.93) | -9.24 (19.79)
  Pain: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Pain: Change at Cycle 14 | -11.66 (19.51) | -9.82 (19.91)
  Pain: Change at Cycle 15: number analyzed (Participants) | 131 | 96
  Pain: Change at Cycle 15 | -11.15 (18.16) | -8.51 (20.94)
  Pain: Change at Cycle 16: number analyzed (Participants) | 116 | 84
  Pain: Change at Cycle 16 | -8.72 (18.02) | -10.52 (21.30)
  Pain: Change at Cycle 17: number analyzed (Participants) | 112 | 73
  Pain: Change at Cycle 17 | -8.88 (18.17) | -9.93 (17.27)
  Pain: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Pain: Change at Cycle 18 | -8.31 (18.33) | -11.19 (18.16)
  Pain: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Pain: Change at Cycle 19 | -6.63 (17.25) | -10.38 (14.51)
  Pain: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Pain: Change at Cycle 20 | -5.72 (19.98) | -10.35 (16.65)
  Pain: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Pain: Change at Cycle 21 | -8.19 (18.27) | -7.55 (16.77)
  Pain: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Pain: Change at Cycle 22 | -9.08 (18.10) | -9.42 (16.72)
  Pain: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Pain: Change at Cycle 23 | -9.66 (20.75) | -8.53 (19.96)
  Pain: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Pain: Change at Cycle 24 | -9.86 (21.56) | -8.76 (15.53)
  Pain: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Pain: Change at Cycle 25 | -10.58 (19.88) | -8.10 (18.69)
  Pain: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Pain: Change at Cycle 26 | -9.01 (17.99) | -9.41 (17.58)
  Pain: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Pain: Change at Cycle 27 | -12.02 (17.28) | -9.23 (14.58)
  Pain: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Pain: Change at Cycle 28 | -11.54 (18.20) | -7.33 (13.46)
  Pain: Change at PT Visit 1: number analyzed (Participants) | 176 | 196
  Pain: Change at PT Visit 1 | -1.70 (23.07) | -2.99 (23.86)
  Pain: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Pain: Change at PT Visit 2 | -7.49 (24.09) | -0.03 (22.04)
  Reflux Symptoms: Cycle 1 (Baseline): number analyzed (Participants) | 367 | 373
  Reflux Symptoms: Cycle 1 (Baseline) | 16.68 (19.03) | 17.34 (18.31)
  Reflux Symptoms: Change at Cycle 2: number analyzed (Participants) | 331 | 333
  Reflux Symptoms: Change at Cycle 2 | -0.13 (16.33) | -1.99 (18.03)
  Reflux Symptoms: Change at Cycle 3: number analyzed (Participants) | 318 | 309
  Reflux Symptoms: Change at Cycle 3 | -0.52 (18.95) | -2.28 (19.53)
  Reflux Symptoms: Change at Cycle 4: number analyzed (Participants) | 295 | 289
  Reflux Symptoms: Change at Cycle 4 | -0.98 (19.18) | -1.90 (19.93)
  Reflux Symptoms: Change at Cycle 5: number analyzed (Participants) | 283 | 285
  Reflux Symptoms: Change at Cycle 5 | -1.92 (18.98) | -1.72 (20.10)
  Reflux Symptoms: Change at Cycle 6: number analyzed (Participants) | 270 | 252
  Reflux Symptoms: Change at Cycle 6 | -2.90 (20.42) | -3.59 (19.04)
  Reflux Symptoms: Change at Cycle 7: number analyzed (Participants) | 239 | 226
  Reflux Symptoms: Change at Cycle 7 | -4.18 (18.36) | -3.20 (20.21)
  Reflux Symptoms: Change at Cycle 8: number analyzed (Participants) | 233 | 213
  Reflux Symptoms: Change at Cycle 8 | -4.96 (19.39) | -5.74 (19.53)
  Reflux Symptoms: Change at Cycle 9: number analyzed (Participants) | 207 | 193
  Reflux Symptoms: Change at Cycle 9 | -5.02 (18.97) | -5.18 (19.81)
  Reflux Symptoms: Change at Cycle 10: number analyzed (Participants) | 186 | 163
  Reflux Symptoms: Change at Cycle 10 | -6.12 (17.81) | -6.48 (18.55)
  Reflux Symptoms: Change at Cycle 11: number analyzed (Participants) | 169 | 153
  Reflux Symptoms: Change at Cycle 11 | -6.44 (18.74) | -6.03 (18.07)
  Reflux Symptoms: Change at Cycle 12: number analyzed (Participants) | 158 | 138
  Reflux Symptoms: Change at Cycle 12 | -4.82 (18.00) | -7.49 (16.99)
  Reflux Symptoms: Change at Cycle 13: number analyzed (Participants) | 141 | 110
  Reflux Symptoms: Change at Cycle 13 | -6.42 (17.09) | -6.77 (18.19)
  Reflux Symptoms: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Reflux Symptoms: Change at Cycle 14 | -5.39 (18.24) | -7.37 (17.45)
  Reflux Symptoms: Change at Cycle 15: number analyzed (Participants) | 131 | 96
  Reflux Symptoms: Change at Cycle 15 | -5.00 (16.66) | -4.98 (18.72)
  Reflux Symptoms: Change at Cycle 16: number analyzed (Participants) | 116 | 84
  Reflux Symptoms: Change at Cycle 16 | -3.07 (18.39) | -4.89 (22.31)
  Reflux Symptoms: Change at Cycle 17: number analyzed (Participants) | 111 | 73
  Reflux Symptoms: Change at Cycle 17 | -3.35 (18.38) | -4.57 (20.44)
  Reflux Symptoms: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Reflux Symptoms: Change at Cycle 18 | -2.94 (18.36) | -6.51 (20.33)
  Reflux Symptoms: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Reflux Symptoms: Change at Cycle 19 | -2.43 (16.38) | -6.15 (18.43)
  Reflux Symptoms: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Reflux Symptoms: Change at Cycle 20 | -1.85 (18.32) | -5.38 (18.63)
  Reflux Symptoms: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Reflux Symptoms: Change at Cycle 21 | -1.83 (18.44) | -4.19 (17.73)
  Reflux Symptoms: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Reflux Symptoms: Change at Cycle 22 | -3.81 (19.30) | -7.00 (19.65)
  Reflux Symptoms: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Reflux Symptoms: Change at Cycle 23 | -5.11 (17.03) | -6.98 (19.70)
  Reflux Symptoms: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Reflux Symptoms: Change at Cycle 24 | -4.07 (19.30) | -7.98 (18.19)
  Reflux Symptoms: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Reflux Symptoms: Change at Cycle 25 | -5.56 (18.86) | -5.71 (16.69)
  Reflux Symptoms: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Reflux Symptoms: Change at Cycle 26 | -4.99 (20.67) | -4.30 (21.98)
  Reflux Symptoms: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Reflux Symptoms: Change at Cycle 27 | -7.75 (20.51) | -6.75 (16.10)
  Reflux Symptoms: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Reflux Symptoms: Change at Cycle 28 | -7.12 (18.64) | -4.44 (11.56)
  Reflux Symptoms: Change at PT Visit 1: number analyzed (Participants) | 176 | 196
  Reflux Symptoms: Change at PT Visit 1 | 0.88 (20.01) | -0.45 (22.92)
  Reflux Symptoms: Change at PT Visit 2: number analyzed (Participants) | 99 | 106
  Reflux Symptoms: Change at PT Visit 2 | 0.56 (18.67) | -1.47 (22.28)
  Taste: Cycle 1 (Baseline): number analyzed (Participants) | 365 | 372
  Taste: Cycle 1 (Baseline) | 13.79 (23.99) | 16.22 (25.49)
  Taste: Change at Cycle 2: number analyzed (Participants) | 328 | 333
  Taste: Change at Cycle 2 | 12.09 (28.78) | 6.61 (26.94)
  Taste: Change at Cycle 3: number analyzed (Participants) | 317 | 307
  Taste: Change at Cycle 3 | 16.72 (32.11) | 9.99 (30.16)
  Taste: Change at Cycle 4: number analyzed (Participants) | 293 | 286
  Taste: Change at Cycle 4 | 18.43 (34.70) | 11.07 (31.93)
  Taste: Change at Cycle 5: number analyzed (Participants) | 282 | 284
  Taste: Change at Cycle 5 | 17.61 (32.93) | 11.85 (30.25)
  Taste: Change at Cycle 6: number analyzed (Participants) | 269 | 251
  Taste: Change at Cycle 6 | 17.97 (31.20) | 11.82 (32.21)
  Taste: Change at Cycle 7: number analyzed (Participants) | 238 | 225
  Taste: Change at Cycle 7 | 16.25 (33.51) | 9.19 (31.09)
  Taste: Change at Cycle 8: number analyzed (Participants) | 232 | 213
  Taste: Change at Cycle 8 | 11.64 (29.81) | 3.29 (28.13)
  Taste: Change at Cycle 9: number analyzed (Participants) | 206 | 193
  Taste: Change at Cycle 9 | 9.22 (28.25) | 1.73 (26.30)
  Taste: Change at Cycle 10: number analyzed (Participants) | 185 | 164
  Taste: Change at Cycle 10 | 7.93 (26.41) | 1.63 (28.79)
  Taste: Change at Cycle 11: number analyzed (Participants) | 168 | 153
  Taste: Change at Cycle 11 | 4.96 (26.72) | 2.61 (26.91)
  Taste: Change at Cycle 12: number analyzed (Participants) | 158 | 138
  Taste: Change at Cycle 12 | 5.27 (24.82) | 0.24 (24.66)
  Taste: Change at Cycle 13: number analyzed (Participants) | 139 | 110
  Taste: Change at Cycle 13 | 4.08 (25.53) | -0.91 (25.33)
  Taste: Change at Cycle 14: number analyzed (Participants) | 136 | 101
  Taste: Change at Cycle 14 | 0.49 (25.66) | -5.28 (24.37)
  Taste: Change at Cycle 15: number analyzed (Participants) | 130 | 96
  Taste: Change at Cycle 15 | 3.08 (24.36) | -1.04 (26.25)
  Taste: Change at Cycle 16: number analyzed (Participants) | 115 | 84
  Taste: Change at Cycle 16 | 5.51 (27.90) | -3.57 (20.71)
  Taste: Change at Cycle 17: number analyzed (Participants) | 111 | 73
  Taste: Change at Cycle 17 | 4.80 (24.96) | -3.65 (23.28)
  Taste: Change at Cycle 18: number analyzed (Participants) | 102 | 70
  Taste: Change at Cycle 18 | 3.59 (23.87) | -4.29 (23.34)
  Taste: Change at Cycle 19: number analyzed (Participants) | 96 | 65
  Taste: Change at Cycle 19 | 3.13 (25.17) | -4.62 (15.45)
  Taste: Change at Cycle 20: number analyzed (Participants) | 84 | 62
  Taste: Change at Cycle 20 | 5.56 (27.78) | -3.76 (18.21)
  Taste: Change at Cycle 21: number analyzed (Participants) | 79 | 53
  Taste: Change at Cycle 21 | 6.33 (27.26) | -5.03 (17.78)
  Taste: Change at Cycle 22: number analyzed (Participants) | 67 | 46
  Taste: Change at Cycle 22 | 9.45 (30.04) | -4.35 (16.64)
  Taste: Change at Cycle 23: number analyzed (Participants) | 63 | 43
  Taste: Change at Cycle 23 | 8.99 (30.06) | 0.00 (23.00)
  Taste: Change at Cycle 24: number analyzed (Participants) | 60 | 39
  Taste: Change at Cycle 24 | 7.78 (28.37) | -5.13 (19.55)
  Taste: Change at Cycle 25: number analyzed (Participants) | 52 | 35
  Taste: Change at Cycle 25 | 3.21 (28.97) | -4.76 (18.33)
  Taste: Change at Cycle 26: number analyzed (Participants) | 49 | 31
  Taste: Change at Cycle 26 | 4.08 (34.45) | -3.23 (21.70)
  Taste: Change at Cycle 27: number analyzed (Participants) | 43 | 28
  Taste: Change at Cycle 27 | 4.65 (29.62) | -3.57 (20.96)
  Taste: Change at Cycle 28: number analyzed (Participants) | 39 | 25
  Taste: Change at Cycle 28 | 3.42 (21.35) | -6.67 (25.46)
  Taste: Change at PT Visit 1: number analyzed (Participants) | 175 | 195
  Taste: Change at PT Visit 1 | 12.76 (34.59) | 9.06 (33.56)
  Taste: Change at PT Visit 2: number analyzed (Participants) | 99 | 105
  Taste: Change at PT Visit 2 | 8.42 (31.35) | 6.67 (28.64)

11. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pertuzumab
Time Frame: Post-dose (0.5 hour after end of 30-60 minutes infusion) on Day 1 of Cycles 1, 2, 4, and 8 (1 cycle = 21 days)
Population: The pharmacokinetic analysis included all participants who were treated with study medication and who had at least one measurable concentration of pertuzumab or trastuzumab. In this analysis, results are reported only for evaluable participants who received pertuzumab.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 374
micrograms per milliliter (μg/mL)
  Cycle 1 | 258 (90.3)
  Cycle 2: number analyzed (Participants) | 346
  Cycle 2 | 288 (83.7)
  Cycle 4: number analyzed (Participants) | 302
  Cycle 4 | 341 (111)
  Cycle 8: number analyzed (Participants) | 106
  Cycle 8 | 371 (127)

12. Secondary Outcome: Cmax of Trastuzumab
Time Frame: Post-dose (0.5 hour after end of 30-60 minutes infusion) on Day 1 of Cycles 1, 2, 4, and 8 (1 cycle = 21 days)
Population: The pharmacokinetic analysis included all participants who were treated with study medication and who had at least one measurable concentration of pertuzumab or trastuzumab. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 372 | 375
μg/mL
  Cycle 1 | 142 (86.8) | 139 (58.6)
  Cycle 2: number analyzed (Participants) | 346 | 354
  Cycle 2 | 120 (46.6) | 120 (44.3)
  Cycle 4: number analyzed (Participants) | 304 | 299
  Cycle 4 | 127 (50.9) | 129 (58.1)
  Cycle 8: number analyzed (Participants) | 115 | 90
  Cycle 8 | 130 (50.8) | 147 (90.2)

13. Secondary Outcome: Minimum Serum Concentration (Cmin) of Pertuzumab
Time Frame: Pre-dose (0-6 hours before infusion) on Day 1 of Cycles 1, 2, 3, 4, 6, and 8 (1 cycle = 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 376
μg/mL
  Cycle 1 | NA (NA) — The Cmin of pertuzumab at Cycle 1 (before first dose) is non-reportable (i.e., lower than quantifiable).
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | 42.4 (24.8)
  Cycle 3: number analyzed (Participants) | 327
  Cycle 3 | 74.0 (40.9)
  Cycle 4: number analyzed (Participants) | 305
  Cycle 4 | 90.4 (42.4)
  Cycle 6: number analyzed (Participants) | 274
  Cycle 6 | 114 (51.8)
  Cycle 8: number analyzed (Participants) | 114
  Cycle 8 | 142 (67.9)

14. Secondary Outcome: Cmin of Trastuzumab
Time Frame: Pre-dose (0-6 hours before infusion) on Day 1 of Cycles 1, 2, 3, 4, 6, and 8 (1 cycle = 21 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 379 | 381
μg/mL
  Cycle 1 | NA (NA) — The Cmin of trastuzumab at Cycle 1 (before first dose) is non-reportable (i.e., lower than quantifiable). | NA (NA) — The Cmin of trastuzumab at Cycle 1 (before first dose) is non-reportable (i.e., lower than quantifiable).
  Cycle 2: number analyzed (Participants) | 345 | 354
  Cycle 2 | 15.4 (11.3) | 17.2 (15.4)
  Cycle 3: number analyzed (Participants) | 328 | 326
  Cycle 3 | 19.9 (13.4) | 20.7 (15.2)
  Cycle 4: number analyzed (Participants) | 305 | 300
  Cycle 4 | 22.9 (12.7) | 24.1 (19.0)
  Cycle 6: number analyzed (Participants) | 274 | 254
  Cycle 6 | 26.3 (14.8) | 29.8 (21.9)
  Cycle 8: number analyzed (Participants) | 114 | 92
  Cycle 8 | 32.7 (15.0) | 37.4 (20.3)

ADVERSE EVENTS:
Time Frame: From Baseline until end of post-treatment follow-up (up to 70 months)
Description: All adverse events (AEs) that occurred during the study and until the post-treatment safety follow-up visit approximately 28 days after last study medication were to be recorded. The safety population included all participants who received any amount of any study medication: those who received any amount of pertuzumab were included in the pertuzumab arm; all other treated participants were included in the placebo arm.
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 299/385 | 318/388
Serious Adverse Events (participants affected / at risk) | 178/385 | 156/388
Other Adverse Events (participants affected / at risk) | 373/385 | 376/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Chemotherapy (N=385) | Placebo + Trastuzumab + Chemotherapy (N=388)
Anaemia (Blood and lymphatic system disorders) | 8 (11) | 16 (19)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect acquired (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Pseudoaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (20) | 20 (22)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastric haemorrhage (Gastrointestinal disorders) | 6 (7) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (9)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 5 (7)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (8) | 13 (17)
Asthenia (General disorders) | 5 (8) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 8 (8) | 9 (9)
Fatigue (General disorders) | 4 (4) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 4 (4) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 3 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Liver abscess (Infections and infestations) | 1 (1) | 2 (2)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (15) | 14 (14)
Pneumonia Klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 8 (8) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 9 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (8) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectosigmoid cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Anticholinergic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (2)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Gastric pneumatosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy bone marrow (Investigations) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Chemotherapy (N=385) | Placebo + Trastuzumab + Chemotherapy (N=388)
Anaemia (Blood and lymphatic system disorders) | 159 (208) | 142 (189)
Leukopenia (Blood and lymphatic system disorders) | 80 (148) | 69 (113)
Neutropenia (Blood and lymphatic system disorders) | 200 (340) | 202 (298)
Thrombocytopenia (Blood and lymphatic system disorders) | 61 (105) | 73 (100)
Abdominal distension (Gastrointestinal disorders) | 25 (36) | 19 (24)
Abdominal pain (Gastrointestinal disorders) | 44 (60) | 51 (59)
Abdominal pain upper (Gastrointestinal disorders) | 28 (33) | 23 (25)
Constipation (Gastrointestinal disorders) | 56 (64) | 84 (107)
Diarrhoea (Gastrointestinal disorders) | 230 (351) | 125 (173)
Dyspepsia (Gastrointestinal disorders) | 24 (27) | 30 (40)
Dysphagia (Gastrointestinal disorders) | 28 (34) | 32 (38)
Nausea (Gastrointestinal disorders) | 224 (314) | 218 (311)
Stomatitis (Gastrointestinal disorders) | 81 (102) | 69 (86)
Vomiting (Gastrointestinal disorders) | 147 (200) | 122 (167)
Asthenia (General disorders) | 59 (83) | 60 (78)
Chills (General disorders) | 37 (37) | 17 (19)
Fatigue (General disorders) | 144 (182) | 123 (166)
Mucosal inflammation (General disorders) | 43 (60) | 34 (40)
Oedema (General disorders) | 20 (33) | 19 (32)
Oedema peripheral (General disorders) | 27 (31) | 33 (36)
Pyrexia (General disorders) | 55 (81) | 60 (69)
Upper respiratory tract infection (Infections and infestations) | 24 (37) | 13 (18)
Infusion related reaction (Injury, poisoning and procedural complications) | 46 (52) | 23 (26)
Blood creatinine increased (Investigations) | 29 (36) | 22 (31)
Creatinine renal clearance decreased (Investigations) | 71 (97) | 50 (65)
Weight decreased (Investigations) | 78 (80) | 49 (51)
Decreased appetite (Metabolism and nutrition disorders) | 172 (243) | 158 (218)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (24) | 21 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 24 (32) | 23 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 74 (98) | 46 (57)
Hypomagnesaemia (Metabolism and nutrition disorders) | 30 (38) | 21 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (19) | 29 (29)
Dizziness (Nervous system disorders) | 31 (35) | 30 (38)
Dysgeusia (Nervous system disorders) | 31 (40) | 27 (27)
Neuropathy peripheral (Nervous system disorders) | 34 (38) | 29 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 29 (37) | 34 (35)
Insomnia (Psychiatric disorders) | 34 (45) | 46 (48)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 21 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 14 (18)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 37 (45)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (25) | 25 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 32 (39) | 18 (21)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 86 (91) | 100 (112)
Pruritus (Skin and subcutaneous tissue disorders) | 38 (51) | 16 (25)
Rash (Skin and subcutaneous tissue disorders) | 27 (30) | 13 (15)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 (17) | 21 (21)
Hypertension (Vascular disorders) | 20 (24) | 21 (21)
Nasopharyngitis (Infections and infestations) | 21 (22) | 18 (24)
Ejection fraction decreased (Investigations) | 20 (24) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.